Clinical Investigation of Visual Acuity in Contact Lens Wearers after Instillation of a Lipid-Based Lubricating Eye Drop

Protocol CR-6371

Version: 4.0

Date: 19 August 2020

Investigational Products: Investigational lipid eye drops and blink® Tears Eye Drops

Key Words: artificial tears, blink® Tears, logMAR Visual Acuity, contact lenses, non-dispensing

#### Statement of Compliance to protocol, GCP and applicable regulatory guidelines:

This trial will be conducted in compliance with the protocol, ISO 14155,<sup>1</sup> the International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP),<sup>2</sup> the Declaration of Helsinki,<sup>3</sup> and all applicable regulatory requirements. This study will be conducted as a non-significant risk device investigation per 21 CFR 812.2 (b) IDE Abbreviated Requirements and per U.S. FDA GUIDANCE FOR INDUSTRY -- Premarket Notification (510[k]) Guidance Document for Contact Lens Care Products dated May 1 1997).

#### **Confidentiality Statement:**

This document contains confidential information, which should not be copied, referred to, released or published without written approval from Johnson & Johnson Vision Care, Inc. The information may not be disclosed to others except to the extent necessary to obtain Institutional Review Board/Independent Ethics Committee approval and informed consent, or as required by International, Federal and State Laws, as applicable. Persons to whom this information is disclosed must be informed that this information is privileged and confidential and that it should not be further disclosed without the written permission of Johnson & Johnson Vision Care, Inc. Any supplemental information that may be added to this document is also confidential and proprietary to Johnson & Johnson Vision Care, Inc. and must be kept in confidence in the same manner as the contents of this document.

| TABLE | E OF CONTENTS | |
|---|---|---|
| PROTO | COL TITLE, NUMBER, VERSION | <i>6</i> |
| SPONS | OR NAME AND ADDRESS | <i>6</i> |
| MEDIC | AL MONITOR | <i>6</i> |
| AUTHO | DRIZED SIGNATURES | 7 |
| CHANG | GE HISTORY | 8 |
| SYNOP | PSIS | 9 |
| COMM | ONLY USED ABBREVIATIONS AND DEFINITIONS OF TERMS | 14 |
| 1. IN | TRODUCTION AND BACKGROUND | 16 |
| 1.1. | Name and Descriptions of Investigational Products | 16 |
| 1.2. | Intended Use of Investigational Products | 16 |
| 1.3. | Summary of Findings from Nonclinical Studies | |
| 1.4. | Summary of Known Risks and Benefits to Human Subjects | 16 |
| 1.5.<br>Study | Relevant Literature References and Prior Clinical Data Relevant to Propose 17 | ed Clinica |
| 2. ST | UDY OBJECTIVES, ENDPOINTS AND HYPOTHESES | 17 |
| 2.1. | Objectives | 17 |
| 2.2. | Endpoints | 17 |
| 2.3. | Hypotheses | 17 |
| 3. TA | ARGETED STUDY POPULATION | 17 |
| 3.1. | General Characteristics | 17 |
| 3.2. | Inclusion Criteria | 18 |
| 3.3. | Exclusion Criteria | 18 |
| 3.4. | Enrollment Strategy | 19 |
| 4. ST | UDY DESIGN AND RATIONALE | 19 |
| 4.1. | Description of Study Design | |
| 4.2. | Study Design Rationale | 19 |
| 4.3. | Enrollment Target and Study Duration | 20 |
| 5. TE | ST ARTICLE ALLOCATION AND MASKING | |
| 5.1. | Test Article Allocation | |
| 5.2. | Masking | |
| 5.3. | Procedures for Maintaining and Breaking the Masking | |
| 6. ST | UDY INTERVENTION | 21 |
| 6.1. | Identity of Test Articles. | 21 |

| 6 | .2. | Ancillary Supplies/Products | . 22 |
|---|---|---|---|
| 6 | 5.3. | Administration of Test Articles | . 22 |
| 6 | .4. | Packaging and Labeling | . 22 |
| 6 | 5.5. | Storage Conditions | . 23 |
| 6 | .6. | Collection and Storage of Samples | . 23 |
| 6 | 5.7. | Accountability of Test Articles | . 23 |
| 7. | STU | UDY EVALUATIONS | . 24 |
| 7 | .1. | Time and Event Schedule | . 24 |
| 7 | .2. | Detailed Study Procedures | . 25 |
| | VIS | SIT 1 | . 25 |
| | FIN | IAL EVALUATION | . 27 |
| 7 | .3. | Unscheduled Visits | . 28 |
| 7 | .4. | Laboratory Procedures | . 29 |
| 8. | SU | BJECTS COMPLETION/WITHDRAWAL | . 29 |
| 8 | .1. | Completion Criteria | . 29 |
| 8 | .2. | Withdrawal/Discontinuation from the Study | . 29 |
| 9. | PR] | E-STUDY AND CONCOMITANT INTERVENTION/MEDICATION | . 30 |
| 9 | .1. | Systemic Medications | . 30 |
| 10. | D | EVIATIONS FROM THE PROTOCOL | . 30 |
| 11. | S | TUDY TERMINATION | . 31 |
| 12. | P | ROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS | . 32 |
| 13. | A | DVERSE EVENTS | . 33 |
| 1 | 3.1. | Definitions and Classifications | . 33 |
| 1 | 3.2. | Assessing Adverse Events | . 35 |
| | 13.2 | 2.1. Causality Assessment | . 35 |
| | 13.2 | 2.2. Severity Assessment | . 36 |
| 1 | 3.3. | Documentation and Follow-Up of Adverse Events | . 36 |
| 1 | 3.4. | Reporting Adverse Events | . 37 |
| | 13.4 | 4.1. Reporting Adverse Events to Sponsor | . 38 |
| | 13.4 | 4.2. Reporting Adverse Events to the Responsible IEC/IRB and Health Authori 38 | ties |
| | 13.4 | 4.3. Event of Special Interest | . 39 |
| 1 | 3.5. | Reporting of Pregnancy | . 39 |
| 14. | S | TATISTICAL METHODS | . 39 |

| 14.1. | General Considerations | 39 |
|---|---|---|
| 14.2. | Sample Size Justification | 39 |
| 14.3. | Analysis Populations | 39 |
| 14.4. | Level of Statistical Significance | 40 |
| 14.5. | Primary Analysis | 40 |
| 14.6. | Secondary Analysis | 40 |
| 14.7. | Other Exploratory Analyses | 40 |
| 14.8. | Interim Analysis | 40 |
| 14.9. | Procedure for Handling Missing Data and Drop-Outs | 40 |
| 14.10. | Procedure for Reporting Deviations from Statistical Plan | 40 |
| 15. D | ATA HANDLING AND RECORD KEEPING/ARCHIVING | 41 |
| 15.1. | Electronic Case Report Form/Data Collection | 41 |
| 15.2. | Subject Record | 41 |
| 15.3 C | linicalTrials.gov | 42 |
| 16. D | ATA MANAGEMENT | 42 |
| 16.1. | Access to Source Data/Document | 42 |
| 16.2. | Confidentiality of Information | 42 |
| 16.3. | Data Quality Assurance | 42 |
| 17. C | LINICAL MONITORING | 43 |
| 18. E | THICAL AND REGULATORY ASPECTS | 43 |
| 18.1. | Study-Specific Design Considerations | 43 |
| 18.2. | Investigator Responsibility | 43 |
| 18.3. | Independent Ethics Committee or Institutional Review Board (IEC/IRB) | 44 |
| 18.4. | Informed Consent | 45 |
| 18.5. | Privacy of Personal Data | 45 |
| 19. S | TUDY RECORD RETENTION | 46 |
| 20. FI | NANCIAL CONSIDERATIONS | 47 |
| 21. PI | JBLICATION | 47 |
| 22. R | EFERENCES | 48 |
| APPENI | DIX A: PATIENT INSTRUCTION GUIDE | 49 |
| APPENI | DIX B: PACKAGE INSERT (APPROVED PRODUCT) | 50 |
| APPENI | <u></u> _ | |
| | SUBJECT REPORTED OCULAR SYMPTOMS | |
| | BIOMICROSCOPY SCALE | 55 |

| DISTANCE AND NEAR VISUAL ACUITY EVALUATION | 61 |
|---------------------------------------------------------|----|
| ETDRS DISTANCE VISUAL ACUITY MEASUREMENT PROCEDURE | 66 |
| VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINA TESTING | |
| APPENDIX D: Guidelines for COVID-19 Risk Mitigation | 76 |
| PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE | 86 |
| TABLE OF CONTENTS Figure 1: Study Flowchart | 13 |
| TABLE OF CONTENTS | |
| Table 1: Lubricating eye drops | 21 |
| Table 2: Ancillary Supplies | |
| Table 3: Time and Events | |

#### PROTOCOL TITLE, NUMBER, VERSION

Title: Clinical Investigation of Visual Acuity in Contact Lens Wearers after Instillation of a

Lipid-Based Eye Drop Protocol Number: CR-6371

Version: 4.0

Date: 19 August 2020

#### SPONSOR NAME AND ADDRESS

Johnson & Johnson Vision Care (JJVC) 7500 Centurion Parkway Jacksonville, FL 32256

#### MEDICAL MONITOR



The Medical Monitor must be notified by the clinical institution/site by e-mail, fax, or telephone within 24 hours of learning of a Serious Adverse Event. The Medical Monitor may be contacted during business hours for adverse event questions. General study related questions should be directed towards your assigned clinical research associate.

The Medical Monitoring Plan is maintained as a separate document and included in the Trial Master File.

#### **AUTHORIZED SIGNATURES**

The signatures below constitutes the approval of this protocol and the attachments and provide the necessary assurances that this trial will be conducted according to all stipulations of the protocol, including all statements regarding confidentiality, and according to local legal and regulatory requirements and applicable U.S. federal regulations, <sup>4</sup> ICH guidelines, <sup>2</sup> ISO 14155, <sup>1</sup> and the Declaration of Helsinki. <sup>3</sup>

| Author/Study<br>Responsible Clinician | See Electronic Signature Report | DATE |
|---|---|---|
| Clinical Operations<br>Manager | See Electronic Signature Report | DATE |
| Biostatistician | See Electronic Signature Report | DATE |
| Data Management | See Electronic Signature Report | DATE |
| Medical Safety Officer | See Electronic Signature Report | DATE |
| Reviewer | Fellow Review is not required | DATE |
| Approver | See Electronic Signature Report | DATE |

#### **CHANGE HISTORY**

| Version | Originator | Description of Change(s) and Section<br>Number(s) Affected | Date |
|---|---|---|---|
| 1.0 | | Original Protocol | 09 September 2019 |
| 2.0 | | Corrected settling time of drops for<br>both treatments, and updated Inclusion<br>criteria for spherical lens wearers | 13 September 2019 |
| 3.0 | | Updated template version, control drop, statistician, and study step clarification | 11 May 2020 |
| 4.0 | | Updated section 13.5, added COVID Risk Mitigation appendix | 19 Aug 2020 |

#### **SYNOPSIS**

| Protocol Title | Clinical Investigation of Visual Acuity in Contact Lens<br>Wearers after Instillation of a Lipid-Based Eye Drop |
|---|---|
| Sponsor | JJVC, 7500 Centurion Parkway, Jacksonville, FL 32256 |
| Clinical Phase | Confirmatory, Phase 1 |
| Trial Registration | This study will be registered on ClinicalTrials.gov based on the following: this study is being conducted after final formulation lock. |
| Test Article(s) | Two lubricating eye drop products: • Investigational lipid eye drops – (Test) • Blink® Tears eye drop (Control) |
| Wear and Replacement Schedules | Not applicable |
| Objectives | The objective of this study is to assess visual acuity after the instillation of a lipid-based eye drop compared to a marketed lubricating eye drop while wearing habitual contact lenses. |
| Study Endpoints | Primary endpoint(s): • Change in logMAR visual acuity after the instillation of the eyedrop. |
| | Other Endpoint(s) • Slit Lamp Findings using FDA scale • Snellen best corrected distance visual acuity • Subject reported ocular symptoms • Adverse Events • Number and reasons for discontinuation will be monitored. |
| Study Design | This is a single visit, randomized, double masked, bilateral, non-dispensing, 2×2 crossover study. |
| Sample Size | Approximately 30 subjects will be enrolled and approximately 25 subjects are targeted to complete the study. |
| Study Duration | The study will last approximately 6 weeks and include a 6-week enrollment period. |
| Anticipated Study Population | Habitual spherical contact lens wearers 18-69 years of age. |

| Eligibility Criteria | Potential subjects must satisfy all of the following criteria to be enrolled in the study: |
|---|---|
| | Inclusion Criteria after Screening: |
| | <ol> <li>The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.</li> <li>Appear able and willing to adhere to the instructions set forth in this clinical protocol.</li> <li>Between 18 and 69 (inclusive) years of age at the time of screening.</li> <li>Subjects must be habitual spherical soft contact lens wearers.</li> </ol> |
| | Inclusion Criteria after Baseline: |
| | 5. Subjects must achieve visual acuity of 20/30 or bette in each eye with their habitual contact lenses. |
| | Potential subjects who meet any of the following criteria wil be excluded from participating in the study: |
| | Exclusion Criteria after Screening: |
| | <ol> <li>Currently pregnant or breast-feeding.</li> <li>Diabetes.</li> <li>Any ocular or systemic allergies or disease which may interfere with the clinical trial (at the discretion of the interfere with the clinical trial).</li> </ol> |
| | <ul><li>investigator).</li><li>4. Any systemic disease, autoimmune disease, or use o medication which may interfere with the clinical tria (at the discretion of the investigator).</li></ul> |
| | 5. Any infectious diseases (e.g. hepatitis, tuberculosis) o a contagious immunosuppressive disease (e.g. HIV) by self-report. |
| | 6. History of any ocular or corneal surgery (e.g. RK PRK, LASIK) |
| | 7. Participation in any pharmaceutical or medical device related clinical trial within 14 days prior to study enrollment. |
| | 8. History of binocular vision abnormality or strabismus 9. Habitual wearers of rigid gas permeable lens within |

the past 3 months

| | <ul> <li>10. Current habitual use of Prescription Medication to treat dry eye or ocular discomfort, ocular steroids, or any medication (RX or OTC) that would interfere with the clinical study (at the discretion of the investigator)</li> <li>11. Employees of investigational clinic (investigator, coordinator, and technician etc) or family members of an employee of the clinical site by self-report.</li> </ul> |
|---|---|
| | Exclusion Criteria after Baseline: |
| | 12. Any Grade 3 or greater biomicroscopy findings (this includes, corneal edema, corneal staining, corneal vascularization, conjunctival injection, tarsal abnormalities, bulbar injection) on the FDA classification scale. |
| | <ul> <li>13. Any active ocular abnormalities/conditions that may interfere with the clinical trial (this includes, but not limited to, chalazia, recurrent styles, pterygium, infection, etc.).</li> <li>14. Any corneal distortion due to previous rigid gas permeable lens wear, surgery or pathology.</li> </ul> |
| | In addition to the above criteria, patients with any allergy or sensitivity to ingredients that this product may contain should not participate in the study (Castor Oil, Polyoxyl 40 Hydrogenated Castor Oil, Sodium Chlorite, Boric Acid, Sodium Borate Decahydrate, Sodium Chloride, Potassium Chloride, Calcium Chloride Dihydrate, Magnesium Chloride Hexahydrate, Polyethylene Glycol 400, Sodium Hyaluronate, Purified Water). |
| Disallowed | Current habitual use of Prescription Medicines to treat dry eye |
| Medications/Interventions | or ocular discomfort, ocular steroids, or any medication (RX or OTC) that would interfere with the clinical study (at the discretion of the investigator). |
| Measurements and | logMAR visual acuity, slit lamp finding using FDA scale, |
| Procedures | Snellen visual acuity, subjective reported ocular symptoms. |
| Microbiology or Other<br>Laboratory Testing | None |

| Study Termination | The occurrence of one or more Unanticipated Adverse Device Effect (UADE), or any serious adverse event (SAE) where relationship to study agent cannot be ruled out, will result in stopping further dispensing investigational product. In the event of a UADE or SAE, the Sponsor Medical Monitor may unmask the treatment regimen of subject(s) and may discuss |
|---|---|
| | this with the Principal Investigator before any further subjects |
| | are enrolled. |
| Ancillary Supplies/ Study- | ScleralFil (Bausch + Lomb), LacriPure (Menicon), |
| Specific Materials Fluorescein (Akorn, Inc.) or other country-specific | |
| | approved by the sponsor. |
| Principal Investigator(s) | A full list of Principal Investigators, clinical sites, and |
| and Study | institutions is kept separately from the Study Protocol and is |
| Institution(s)/Site(s) included in the study Trial Master File. | |

Figure 1: Study Flowchart



#### COMMONLY USED ABBREVIATIONS AND DEFINITIONS OF TERMS

ADD Plus Power Required For Near Use

ADE Adverse Device Effect

AE Adverse Event/Adverse Experience
BCVA Best Corrected Visual Acuity

BSCVA Best Spectacle Corrected Visual Acuity

CFR Code of Federal Regulations
CLUE Contact Lens User Experience

COAS Complete Ophthalmic Analysis System

COM Clinical Operations Manager CRA Clinical Research Associate

CRF Case Report Form

CRO Contract Research Organization

CT Center Thickness

D Diopter

DMC Data Monitoring Committee eCRF Electronic Case Report Form EDC Electronic Data Capture

ETDRS Early Treatment Diabetic Retinopathy Study

FDA Food and Drug Administration

GCP Good Clinical Practice

HIPAA Health Insurance Portability and Accountability Act

IB Investigator's Brochure ICF Informed Consent Form

ICH International Conference on Harmonization

IDE Investigational Device Exemption IEC Independent Ethics Committee IRB Institutional Review Board

ISO International Organization for Standardization

ITT Intent-to-Treat

JJVC Johnson & Johnson Vision Care, Inc.

LC Limbus Center

LogMAR Logarithm of Minimal Angle of Resolution MedDRA<sup>©</sup> Medical Dictionary for Regulatory Activities

MOP Manual of Procedures

NIH National Institutes of Health

OD Right Eye

OHRP Office for Human Research Protections
OHSR Office for Human Subjects Research

OS Left Eye

OTC Over the Counter

OU Both Eyes

PD Protocol Deviation

PHI Protected Health Information

PI Principal Investigator
PIG Patient Instruction Guide
PQC Product Quality Complaint
PRO Patient Reported Outcome

QA Quality Assurance
QC Quality Control
RX Prescription

SAE Serious Adverse Event/Serious Adverse Experience

SAP Statistical Analysis Plan SAS Statistical Analysis System

SD Standard Deviation

SOP Standard Operating Procedure

UADE Unanticipated Adverse Device Effect

USADE Unanticipated Serious Adverse Device Effect

VA Visual Acuity

#### 1. INTRODUCTION AND BACKGROUND

Lubricating eye drops are often used to treat symptoms of ocular dryness and discomfort. Most of the major lubricating eye drop manufacturing companies have some type of lipid product to address lipid deficient tear films, however JJV CEH does not currently have a lipid-like lubricating drop in our portfolio.

This study will be conducted at one clinical site in the United States and will include one investigational lipid eye drop ( ) and one marketed lubricating eye drop (blink® Tears). By developing a lipid-like drop addition to the CEH portfolio it would continue to support JJV Eye Health Mission.

#### 1.1. Name and Descriptions of Investigational Products

The products used in this clinical study are listed below:

- Investigational lipid eye drops (Test)
- Blink® Tears (Control)

#### 1.2. Intended Use of Investigational Products

One of the products is an investigational, preserved lipid drop, and the other product is a marketed eye drop in the U.S. and the EU, available over the counter (without a prescription). Subjects will be required to use the 1 drop in both eyes.

The intended use of the study lubricating drops is treatment of subjects with symptoms of ocular dryness.

#### 1.3. Summary of Findings from Nonclinical Studies

All previous pre-clinical findings were deemed satisfactory prior to proceeding with clinical trials on humans. For the most comprehensive nonclinical information regarding Investigational lipid eye drops refer to the latest version of the Investigator's Brochure.

#### 1.4. Summary of Known Risks and Benefits to Human Subjects

The following risks/adverse events can be associated with using lubricating eye drops and contact lenses, in general:

- There may be less comfort than when the drop was first placed on the eye.
- The eyes may burn, sting and/or itch.
- There may be a feeling of something in the eye (foreign body, scratched area).
- There may be the potential for some temporary impairment due to peripheral infiltrates, peripheral corneal ulcers and corneal erosion.
- There may be the potential for other physiological observations, such as local or generalized edema, corneal neovascularization, corneal staining, injection, tarsal abnormalities, iritis and conjunctivitis, some of which are clinically acceptable in low amounts.
- There may be excessive watering, unusual eye secretions, or redness of the eye.

• Poor visual acuity, blurred vision, rainbows or halos around objects, photo-phobia, or dry eyes may also occur if the drops are used continuously or for too long a time.

There is no direct benefit to the subject for participating in the study, although they will be able to try out new lubricating eye drops. The information from this study will aid if the further development and design of new lubricating eye drops.

For the most comprehensive clinical information regarding the lubricating eye drops refer to the package inserts (Appendix B) and the latest version of the Investigator Brochure.

## 1.5. Relevant Literature References and Prior Clinical Data Relevant to Proposed Clinical Study

Refer to the Investigator's Brochure and package insert (APPENDIX B).

#### 2. STUDY OBJECTIVES, ENDPOINTS AND HYPOTHESES

#### 2.1. Objectives

The objective of this study is to assess visual acuity after the instillation of a lipid-based eye drop compared to a marketed lubricating eye drop while wearing habitual contact lenses.

#### 2.2. Endpoints

Primary Endpoint

Change in logMAR visual acuity after the instillation of a lipid-based eye drop.

Other Exploratory Endpoints

- Slit Lamp Findings using FDA scale
- Snellen best corrected distance visual acuity
- Subject reported ocular symptom
- Adverse Events
- Number and reasons for discontinuation will be monitored.

#### 2.3. Hypotheses

This is a descriptive feasibility study to assess the change in logMAR visual acuity after the instillation of a lipid-based eye drop. No formal hypothesis testing will be performed.

#### 3. TARGETED STUDY POPULATION

#### 3.1. General Characteristics

Habitual contact lens wearers 18-69 years of age.


#### 3.2. Inclusion Criteria

Potential subjects must satisfy all of the following criteria to be enrolled in the study:

Inclusion Criteria after Screening:

- 1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
- 2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
- 3. Between 18 and 69 (inclusive) years of age at the time of screening.
- 4. Subjects must be habitual spherical soft contact lens wearers.

#### Inclusion Criteria after Baseline:

5. Subjects must achieve visual acuity of 20/30 or better in each eye with their habitual contact lenses.

#### 3.3. Exclusion Criteria

Potential subjects who meet any of the following criteria will be excluded from participating in the study:

Exclusion Criteria after Screening:

- 1. Currently pregnant or breast-feeding.
- 2. Diabetes.
- 3. Any ocular or systemic allergies or disease which may interfere with the clinical trial (at the discretion of the investigator).
- 4. Any systemic disease, autoimmune disease, or use of medication which may interfere with the clinical trial (at the discretion of the investigator).
- 5. Any infectious diseases (e.g. hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g. HIV), by self-report.
- 6. History of any ocular or corneal surgery (e.g. RK, PRK, LASIK)
- 7. Participation in any pharmaceutical or medical device related clinical trial within 14 days prior to study enrollment.
- 8. History of binocular vision abnormality or strabismus.
- 9. Habitual wearers of rigid gas permeable lens within the past 3 months
- 10. Current habitual use of Prescription Medication to treat dry eye or ocular discomfort, ocular steroids, or any medication (RX or OTC) that would interfere with the clinical study (at the discretion of the investigator)
- 11. Employees of investigational clinic (investigator, coordinator, and technician etc) or family members of an employee of the clinical site by self-report.

#### Exclusion Criteria after Baseline:

- 12. Any Grade 3 or greater biomicroscopy findings (this includes, corneal edema, corneal staining, corneal vascularization, conjunctival injection, tarsal abnormalities, bulbar injection) on the FDA classification scale.
- 13. Any active ocular abnormalities/conditions that may interfere with the clinical trial (this includes, but not limited to, chalazia, recurrent styles, pterygium, infection, etc.).
- 14. Any corneal distortion due to previous rigid gas permeable lens wear, surgery or pathology.

In addition to the above criteria, patients with any allergy or sensitivity to ingredients that this product may contain should not participate in the study (Castor Oil, Polyoxyl 40 Hydrogenated Castor Oil, Sodium Chlorite, Boric Acid, Sodium Borate Decahydrate, Sodium Chloride, Potassium Chloride, Calcium Chloride Dihydrate, Magnesium Chloride Hexahydrate, Polyethylene Glycol 400, Sodium Hyaluronate, Purified Water).

#### 3.4. Enrollment Strategy

Study subjects will be recruited from the Institution/clinical site's subject database and/or utilizing Independent Ethics Committee (IEC) or Institutional Review Board (IRB) approved materials.

#### 4. STUDY DESIGN AND RATIONALE

#### 4.1. Description of Study Design

This is a single visit, randomized, double-masked, bilateral, controlled, 2×2 crossover study. Approximately 30 subjects will be screened and randomly assigned to either Test or Control group. The goal is for a sample size of 25 after subjects who withdraw or are lost-to-follow-up.

At Visit 1, subjects will be consented and screened for inclusion/exclusion criteria. Baseline logMAR visual acuity will be measured in their habitual contact lenses. If a subject is found to meet all eligibility criteria, the first lubricating eye drops will be instilled based on the randomization scheme; otherwise, the subject will be discontinued from the study. Three minutes and ten minutes after OD drop instillation logMAR visual acuity will be measured. There will then be a 90 minutes washout period. After the washout, the second artificial tear eye drop will be instilled. Three minutes and ten minutes after instillation logMAR visual acuity will be measured. The subject will then complete the final evaluation.

#### 4.2. Study Design Rationale

Randomized, double masked, controlled designs are the gold standard to perform scientifically sound evaluations of the intervention by reducing bias associated with the conduct and interpretation of a clinical trial and avoiding confounding from other factors. Crossover study design was chosen to allow more efficient comparison of the test articles.

#### 4.3. Enrollment Target and Study Duration

Up to 30 subjects will be enrolled (informed consent signed) and randomized from up to 2 sites in the US. The goal is for a sample size of 25 subjects after subjects who withdraw or are lost to follow-up.

The Investigator is responsible for ensuring that all subjects entering the study conform to subject selection criteria.

#### 5. TEST ARTICLE ALLOCATION AND MASKING

#### 5.1. Test Article Allocation

Subjects will be randomly assigned to one of two unique sequence groups to bilaterally receive two different test articles one at a time over two study periods. The randomization scheme will be generated using the PROC PLAN procedure from the Statistical Analysis System (SAS) Software version 9.4 or higher.<sup>7</sup>

The study site will follow the randomization scheme provided and will complete enrollment according to the randomization list and will not pre-select or assign subjects. The assignment of the subjects must be performed at the first baseline visit (Visit 1). The following must have occurred prior to randomization:

- Informed consent has been obtained
- Subject meets all the inclusion / exclusion criteria
- Subject history and baseline information has been collected

#### 5.2. Masking

This is a double masked study where subjects and the investigators are masked to the identity of the eye drops during the study period. Every attempt will be made to keep the other clinical trial personnel involved in the study (e.g., Data management, Biostatistician) unaware of the identity of the test articles.

The identity of the investigational products will be masked by over labeling the eye drop bottles with a label containing the study number, expiration date and the randomization codes. Only the personnel involved in the over labeling and the unmasked Statistician generating the randomization scheme will have access to the decode information translating the randomization codes into Test and Control eye drops. The medical monitor will also have access to the decode information in case breaking the mask is necessary for the urgent medical treatment of a subject.

#### 5.3. Procedures for Maintaining and Breaking the Masking

Under normal circumstances, the mask should not be broken until all subjects have completed the study and the database is finalized. Otherwise, the mask should be broken only if specific emergency treatment/course of action would be dictated by knowing the treatment status of the

subject. In such cases, the Investigator may, in an emergency, contact the medical monitor. In the event the mask is broken, the Sponsor must be informed as soon as possible. The date, time, and reason for the unmasking must be documented in the subject record. The Investigator is also advised not to reveal the study treatment assignment to the clinical site or Sponsor personnel.

When dispensing test articles, the following steps should be followed to maintain randomization codes:

- 1. Investigator or designee (documented on the Delegation Log) will consult the randomization scheme to obtain the test article assignment for that subject prior to dispensing
- 2. Investigator or designee will record the subject's number on the appropriate line of the randomization scheme
- 3. Investigator or designee will pull the appropriate test articles from the study supply. All test articles that are opened, whether dispensed (placed/fit on eye or dispensed outside the clinical site) or not, must be recorded on the Test Article Accountability Log in the "Dispensed" section.

#### 6. STUDY INTERVENTION

#### **6.1.** Identity of Test Articles

Table 1: Lubricating eye drops

| | Test | Control |
|---|---|---|
| Solution | Investigational lipid eye drops | Blink® Tears |
| Name/Description | | |
| Manufacturer | Johnson & Johnson Vision, Inc | Johnson & Johnson Vision, Inc |
| Ingredients | Castor Oil, Polyoxyl 40 | See package insert |
| | Hydrogenated Castor Oil, | |
| | Sodium Chlorite, Boric Acid, | |
| | Sodium Borate Decahydrate, | |
| | Sodium Chloride, Potassium | |
| | Chloride, Calcium Chloride | |
| | Dihydrate, Magnesium Chloride | |
| | Hexahydrate, Polyethylene | |
| | Glycol 400, Sodium | |
| | Hyaluronate, Purified Water | |
| Packaging Form | Over-Labeled | Over-Labeled |

#### 6.2. Ancillary Supplies/Products

ScleralFil (Bausch + Lomb) or LacriPure (Menicon) or other country-specific alternative approved by the sponsor may be used to rinse the eye following instillation of Sodium fluorescein dye.

Table 1: Ancillary Supplies

| | | Solution | |
|---|---|---|---|
| Solution Name/Description | ScleralFil (or<br>other sponsor-<br>approved<br>product) | Lacripure (or<br>other sponsor-<br>approved<br>product) | Fluorescein (or<br>other sponsor-<br>approved<br>product) |
| Manufacturer | Bausch + Lomb | Menicon | Akorn, Inc |
| Preservative | None | None | None |
| Other distinguishing items (dye, packaging, approval status, etc.) | NA | NA | D&C Yellow No.<br>8, 0.6 mg |

Sodium fluorescein dye will be used for biomicroscopy, as needed. Sterile, preservative-free, saline may be used in this clinical study to rinse each eye.

#### 6.3. Administration of Test Articles

Test articles will be administered to subjects meeting all eligibility requirements set forth in this clinical protocol. Lost or damaged test articles will not be replaced at the discretion of the Investigator and/or the Sponsor.

#### 6.4. Packaging and Labeling

The test articles will be packaged in bottles as the primary packaging. The test article will be over-labeled to mask the subject to the identity. The test articles will be in investigational cartons sealed with a tamper evident seal, commercial cartons, or in plastic bags as the secondary packaging form. The labels for the primary and secondary packages will contain the following message, in accordance with JJV over-labeling procedures for masked studies involving marketed products: "For Use in Clinical Study CR-6371, Eye Drops. CAUTION – For Investigational Use Only." The labels will also contain the product code, lot number, expiration date and the clinical study number.



#### 6.5. Storage Conditions

Test articles will be maintained at ambient temperatures at the clinical site. Test articles must be kept under secure conditions.

#### 6.6. Collection and Storage of Samples

When possible, any test article associated with an Adverse Event and/or a Product Quality Complaint must be retained pending directions from the sponsor for potential return to JJVC.

#### 6.7. Accountability of Test Articles

JJVC will provide the Investigator with sufficient quantities of study articles and supplies to complete the investigation. The Investigator is asked to retain all lens shipment documentation for the test article accountability records.

Test articles must be kept in a locked storage cabinet, accessible only to those assigned by the Investigator for dispensing. The Investigator may delegate this activity to authorized study site personnel listed on the Site Delegation Log. All test articles must be accounted. This includes:

- 1. What was dispensed to the subject for in-office use.
- What was returned to the Investigator unused, including expired or malfunctioning product.
- 3. The number and reason for unplanned replacements.

The Investigator will collect all unused test articles from the subjects at the end of the subject's participation. Subject returned unused test articles must be separated from the clinical study inventory of un-dispensed test articles and must be labeled with the subject number and date of return. Following final reconciliation of test articles by the monitor, the Investigator or monitor will return all unused test articles to JJVC.

If there is a discrepancy between the shipment documents and the contents, contact the study monitor immediately.

#### 7. STUDY EVALUATIONS

#### 7.1. Time and Event Schedule

Table 2: Time and Events

| Visit Information Time Point | Visit 1<br>Baseline,<br>dispense<br>drop<br>Day 0 |
|---|---|
| Estimated Visit<br>Duration | 3 hours |
| Study Informed Consent | X |
| Inclusion/Exclusion<br>Screening Criteria | X |
| Demographics | X |
| Medical History & medication review | X |
| Entrance Snellen VA | X |
| Biomicroscopy | X |
| Eligibility | X |
| Randomization | X |
| Baseline logMAR | X |
| Instillation of drop #1 | X |
| Ocular symptoms | X |
| 3-minute post drop #1<br>logMAR | X |
| 10-minute post drop #1<br>logMAR | X |
| 90-minute washout | X |
| Instillation of drop #2 | X |
| Ocular symptoms | X |
| 3-minute post drop #2<br>logMAR | X |
| 10-minute post drop #2<br>logMAR | X |
| Exit Slit-lamp | X |
| Exit Snellen VA | X |
| Final Evaluation | X |

### 7.2. Detailed Study Procedures

VISIT 1
Subjects should attend the Visit 1 while wearing their habitual contact lenses.

| Visit 1: Screening | | |
|---|---|---|
| Step | Procedure | Details |
| 1.1 | Statement of<br>Informed Consent | Each subject must read, understand, and sign the Statement of Informed Consent before being enrolled into the study. The Principal Investigator or his/her designee conducting the informed consent discussion must also sign the consent form. NOTE: The subject must be provided a |
| 1.2 | Demographics | Record the subject's date of birth, gender, race and ethnicity. |
| 1.3 | Medical History and<br>Concomitant<br>Medications | Questions regarding the subjects' medical history and concomitant medications. |
| 1.4 | Habitual Lenses | Questions regarding the subject's habitual lens type and parameters. |
| 1.5 | Wear time and<br>comfortable wear<br>time with Habitual<br>Lenses | Record the subject's wear time and comfortable wear time with their habitual contact lenses. |
| 1.6 | Eligibility after<br>Screening | All responses to Screening Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria must be answered "no" for the subject to be considered eligible. If subject is deemed to be ineligible after screening, proceed to Final Evaluation and complete Subject Disposition. Refraction and Biomicroscopy forms are not required. |

| | Visit 1: Baseline | | |
|---|---|---|---|
| Step | Procedure | Details | -, |
| 1.7 | Entrance Visual<br>Acuity | Record the distance Snellen visual acuity (OD, OS, and OU) to the nearest letter with their habitual contact lens correction in place. Subjects must read the smallest line until at least 50% of the letters are read incorrectly. | |

| | Visit 1: Baseline | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 1.8 | Baseline SROS | Subjects will respond to a verbal open-ended symptoms questionnaire. | |
| 1.9 | Remove habitual<br>Contact lenses | Remove habitual contact lenses and store in a case with non-preserved saline. | |
| 1.10 | Slit Lamp<br>Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings and determine eligibility. If any of these slit lamp findings are grade 3 or higher, the subject may not continue at this time, but may return up to one additional time to determine eligibility. If discontinued a final examination must be completed. | |
| | | If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. | |
| 1.11 | Eligibility after<br>Baseline | All responses to Inclusion Criteria questions must be answered "yes" and all responses to Exclusion Criteria questions must be answered "no" for the subject to be considered eligible. If subject is deemed to be ineligible after baseline, proceed to Final Evaluation and complete all forms. | |
| 1.12 | Reinsert habitual lenses | Habitual lenses will be reinserted | |
| 1.13 | Settling time | Allow habitual lenses 5 minutes to settle. | (S) |
| 1.14 | Baseline Distance<br>ETDRS LogMAR<br>Visual Acuity | Under high illumination and high chart luminance, record the distance (4 meter) ETDRS low contrast visual acuity OD (LC1) and OS (LC2). | |

| | Visit 1: Treatment 1 | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 1.15 | Drop Selection | Assign the study drop based on the randomization scheme. | Tu 50 |
| 1.16 | Drop Instillation | The Investigator or technician will instill 1 drop in the right eye. Wait 1 minute and then instill 1 drop in the left eye. | |

| | Visit 1: Treatment 1 | |
|---|---|---|
| Step | Procedure | Details |
| 1.17 | Ocular Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire. |
| 1.18 | Drop Settling | Allow the drop to settle for 3 minutes (from OD drop). |
| 1.19 | 3-minute Distance<br>ETDRS LogMAR<br>Visual Acuity (from<br>OD drop time) | Under high illumination and high chart luminance, record the distance (4 meter) ETDRS low contrast visual acuity OD (LC3) and OS (LC4). |
| 1.20 | | Under high illumination and high chart luminance, record the distance (4 meter) ETDRS low contrast visual acuity OD (LC1) and OS (LC2). |
| 1.21 | Drop Wash out | Allow a washout of at least 90 minutes before continuing to the second eye drop (subject continue to wear habitual contact lenses during this time). |

| | Visit 1: Treatment 2 | | |
|---|---|---|---|
| Step | Procedure | Details | |
| 1.22 | Drop Instillation | The Investigator or technician will instill 1 | de 10 |
| | 02652 | drop in right eye, wait 1 minute and then | |
| | | instill 1 drop in the left eye. | |
| 1.23 | Ocular Symptoms | Subjects will respond to a verbal open-ended | |
| | | symptoms questionnaire. | - |
| 1.24 | Drop Settling | Allow the drop to settle for 3 minutes (from | |
| | | OD drop time). | |
| 1.25 | 3-minute Distance | Under high illumination and high chart | |
| | ETDRS LogMAR | luminance, record the distance (4 meter) | |
| | Visual Acuity (from | ETDRS low contrast visual acuity | |
| | OD drop time) | OD (LC3) and OS (LC4). | |
| 1.26 | 10-minute Distance | Under high illumination and high chart | |
| | ETDRS LogMAR | luminance, record the distance (4 meter) | |
| | Visual Acuity (from | ETDRS low contrast visual acuity | |
| | OD drop time) | OD (LC1) and OS (LC2). | |
| 1.27 | Remove habitual | Remove habitual contact lenses and store in a | |
| | Contact lenses | case with non-preserved saline. | |

#### FINAL EVALUATION

The final evaluation will ordinarily take place immediately following the last scheduled follow-up visit per the study protocol. It may also take place at any point the subject discontinues the study or is terminated from the study.

| | Final Evaluation | |
|---|---|---|
| Step | Procedure | Details |
| F.1 | Final Exam Form | Indicate if the subject completed the study successfully. If subject discontinued from the study, indicate the reason. |
| F.2 | Exit Slit Lamp<br>Biomicroscopy | FDA Slit Lamp Classification Scale will be used to grade the findings and determine eligibility. If the clearance of the fluorescein needs to be expedited, preservative-free rewetting drops or saline may be instilled. |
| F.3 | Exit Visual Acuity | Record the distance Snellen visual acuity (OD, OS, and OU) to the nearest letter with their habitual contact lens correction in place. Subjects must read the smallest line until at least 50% of the letters are read incorrectly. |

#### 7.3. Unscheduled Visits

If, during the investigation, a subject requires an unscheduled visit to the clinical site, the following information will be collected at a minimum:

- Chief complaint prompting the visit. If the reason is an adverse event, the applicable eCRF for the adverse event must be completed and subject record completed as appropriate.
- Date and time of the visit and all procedures completed at the unscheduled visit.
- Review of adverse event and concomitant medications.
- Documentation of any test article dispensed or collected from the subject, if applicable.
- Slit lamp findings (using the Slit Lamp Classification Scale).

If the Investigator withdraws a subject from the study, the final study visit case report forms must be completed indicating the reason(s) why the subject was withdrawn. The subject record must be completed documenting the date and primary reason for withdrawal and the study CRA notified.

Any ocular and non-ocular Adverse Events that are ongoing at the time of the study visit will be followed by the Investigator, within licensure, until they have resolved, returned to pretreatment status, stabilized, or been satisfactorily explained. If further treatment i.e., beyond licensure is required, the subject will be referred to the appropriate health care provider.

The following information may be collected during an unscheduled visit, as applicable depending on the chief complaint/reason for visit.

| | Unscheduled Visit | | |
|---|---|---|---|
| Step | Procedure | Details | |
| U.1 | Chief Complaints | Record the subject's chief complaints for | |
| | | reasons for the unscheduled visit. | |
| U.2 | Adverse Events and | Review any changes to the subject's medical | |
| | Concomitant | history or concomitant medications from the | |
| | Medications Review | previous study visit. Record any changes, and | |
| | | any adverse events. | |
| U.3 | Entrance VA | Record the entrance distance visual acuity | |
| | | (OD, OS and OU) to the nearest letter. | |
| U.4 | Subjective Sphero- | Perform bare-eye subjective spherocylindrical | |
| | cylindrical | refraction with a phoropter (adopt the | |
| | Refraction | maximum plus to maximum visual acuity | |
| | | (MPMVA) approach and use the duo-chrome | |
| | | test for binocular balancing) and record the | |
| | | best corrected distance visual acuity to the | |
| | | nearest letter (OD, OS, and OU). | |
| U.5 | Slit Lamp | FDA Slit Lamp Classification Scale will be | |
| | Biomicroscopy | used to grade the findings. If the clearance of | |
| | | the fluorescein needs to be expedited, | |
| | | preservative-free rewetting drops may be | |
| | | instilled. | <u> </u> |
| U.6 | Exit Visual Acuity | Record the subject's exit distance visual | |
| | | acuity (OD, OS, and OU) to the nearest letter. | |

#### 7.4. Laboratory Procedures

Not applicable.

#### 8. SUBJECTS COMPLETION/WITHDRAWAL

#### 8.1. Completion Criteria

Subjects are considered to have completed the study if they:

- Provided informed consent;
- They are eligible;
- Completed all study visits;
  - Have not withdrawn/discontinued from the study for any reason described in Section 8.2

#### 8.2. Withdrawal/Discontinuation from the Study

A subject will be withdrawn from the study for any of the following reasons:

- Subject death during the study period
- Subject withdrawal of consent
- Subject not compliant to the study protocol including drop usage schedule

- Subject lost to follow-up
- Subject no longer meets eligibility criteria (e.g. the subject becomes pregnant)
- Subject develops significant or serious adverse events causing discontinuation of study drop
- Subjects who have experienced a Corneal Infiltrative Event (CIE)
- Investigator's clinical judgment regarding the subject safety reasons (that it is in the best interest of the subject to stop treatment)
- Subject not successfully dispensed due to lack of efficacy or safety.

For discontinued subjects, the Investigator will:

- Complete the current visit (scheduled or unscheduled)
- Complete the Final Evaluation, indicating the reason that the subject was discontinued from the study

An additional subject may be enrolled if a subject discontinues from the study prematurely.

In cases where a subject is lost to follow-up, every possible effort must be made to contact the subject and determine the reason for discontinuation/withdrawal. The measures taken to follow up must be documented including two written attempts and a certified letter (or equivalent) as the final attempt.

#### 9. PRE-STUDY AND CONCOMITANT INTERVENTION/MEDICATION

Concomitant medications will be documented during screening and updated during the study. Disallowed medications for this study include: Current habitual use of Prescription Only Medicines for dry eye or ocular discomfort, ocular steroids, or any medication (RX or OTC) that would interfere with the clinical study (at the discretion of the investigator).

#### 9.1. Systemic Medications

Due to the nature of the study and endpoints being assessed, medications will be allowed provided they did not interfere with contact lens wear, which will be at the discretion of the investigator.

#### 10. DEVIATIONS FROM THE PROTOCOL

Investigator will notify study sponsor upon identification of a protocol deviation. Protocol deviations must be reported to the sponsor within 24 hours after discovery of the protocol deviation. The Investigator will report deviations per IRB/IEC requirements. All deviations will be tracked and corrective actions implemented as appropriate.


If it becomes necessary for the Investigator to implement a deviation in order to eliminate an immediate hazard to the trial subject, the Investigator may implement the deviation immediately without notification to the sponsor. Within 24 hours after the implemented deviation, the Investigator must notify and provide the rationale to the Sponsor and, as required, the IEC/IRB.

If the deviation potentially impacts the safety of patient or changes the technical integrity of the study then it must be reported to IEC/IRB. This is a "Major Deviation".

Minor deviations have no substantive effect on patient safety or technical integrity of the study. They are often logistical in nature. The informed consent must also not be contradicted by the deviation.

Visual performance assessments started at 2 minutes, or between 4 and 5 minutes after OD drop insertion will be considered minor deviations. Visual performance assessments started 1 minute or less, or 6 minutes or more after OD drop insertion will be considered major deviations for the 3-minute LogMAR procedure (Steps 1.19 and 1.25).

Visual performance assessments started at 8 minutes, or between 11 and 12 minutes after OD drop insertion will be considered minor deviations. Assessments started 7 minutes or less, or 13 minutes or more after OD drop insertion will be considered major deviations for the 10-minute LogMAR procedure (Steps 1.20 and 1.26).

Protocol waivers are prohibited.

#### 11. STUDY TERMINATION

The occurrence of one or more Unanticipated Serious Adverse Device Effect (USADE), or any SAE where the relationship to study agent cannot be ruled out, may result in stopping further dispensing of test article. In the event of a USADE or SAE, the Sponsor may unmask the treatment regimen for the subject(s) and will discuss this with the Investigator before any further subjects are enrolled.

The Sponsor will determine when a study will be stopped. The Principal Investigator always has the discretion to initiate stopping the study based on patient safety or if information indicates the study's results are compromised.

JJVC reserves the right to terminate the study at any time for any reason. Additionally, the IEC/IRB reserves the right to terminate the study if an unreasonable risk is determined. The study can be terminated by the Principal Investigator at the individual clinical site due to specific clinical observations, if in their opinion, after a discussion with JJVC, it is determined that it would be unwise to continue at the clinical site.

JJVC (and the IEC/IRB and DMC, if applicable) will evaluate all adverse events. If it is determined that an adverse event presents an unreasonable risk, the investigation, or that part of the investigation presenting the risk, will be terminated as soon as possible.

Should the study be terminated (either prematurely or as scheduled), the Investigator will notify the IEC/IRB and Regulatory Authority as required by local regulatory requirements.

#### 12. PROCEDURE FOR HANDLING PRODUCT QUALITY COMPLAINTS

A Product Quality Complaint (PQC) refers to any written, electronic, or oral communication that alleges deficiencies related to the identity, quality, durability, reliability, safety, effectiveness or performance of test articles after they have been released for clinical trial use.

Potential complaints may come from a variety of sources including but not limited to subjects, clinical research associates (CRA), clinical operations managers (COM), medical monitors, and site personnel, etc. The following are not considered product quality complaints:

- Subject satisfaction inquiries reported via "Subjective Questionnaires" and "Patient Reported Outcomes (PRO)."
- Clinical test articles that are stored improperly or damaged after receipt at the investigational site.
- Test article replacements that occur due to missed drops.
- Damage deemed by clinicians or clinical staff to be caused by handling by the user, and not indicative of a quality deficiency, only in situations where there is no deficiency alleged by the subject.

Within 24 hours of site personnel becoming aware that a PQC has occurred, the PQC must be recorded in the EDC system, which will trigger an automatic email notification to the appropriate COM/CRA and Clinical QA representative. In cases where the EDC system in use is not configured to send automatic notifications or when an EDC system is not used, the COM/CRA is responsible for notifying Clinical QA upon discovery that a PQC has occurred.

Upon receipt of the EDC notification, the COM/CRA will contact the study site to collect additional information which will include:

- Date the complaint was received/recorded in the EDC System (Date of Sponsor Awareness).
- Who received the complaint.
- Study number.
- Clinical site information (contact name, site ID, telephone number).
- Lot number(s).
- Unique Subject Identifier(s).
- Indication of who first observed complaint (site personnel or subject).
- OD/OS indication, along with whether the lens was inserted.
- Any related AE number if applicable.
- Detailed complaint description (scheduled/unscheduled visit, wear time, symptoms, resolution of symptoms, etc.).
- Eye Care Provider objective (slit lamp) findings if applicable.

Confirmation of product availability for return (and tracking information, if available),
 or rationale if product is not available for return

Once a complaint is received, it will be assessed by the COM, CRA, or trained site personnel to determine if it is an Adverse Event/Serious Adverse Event (AE/SAE). If the complaint results in an AE/SAE, the COM/CRA, or trained site personnel will follow Section 13 of this protocol. If the AE/SAE was potentially the result of a product quality related deficiency, these procedures also applies and will be executed in parallel.

In some cases, a PQC form may be generated in EDC by the site in error. In this event, the PQC forms will be marked "Intentionally Left Blank" or "ILB". Justification for ILB must be documented.

#### 13. ADVERSE EVENTS

#### 13.1. Definitions and Classifications

**Adverse Event (AE)** – An AE is "any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in subjects, users or other persons, whether or not related to the investigational medical device. This definition includes events related to the investigational medical device or the comparator, and to the procedures involved. For users or other persons, this definition is restricted to events related to investigational medical devices<sup>1</sup>

An AE includes any condition (including a pre-existing condition) that:

- 1. Was not present prior to the study, but appeared or reappeared following initiation of the study.
- 2. Was present prior to the study, but worsened during the study. This would include any condition resulting from concomitant illnesses, reactions to concomitant medications, or progression of disease states.
- 3. Pregnancy must be documented as an adverse event and must be reported to the clinical monitor and to the Sponsor immediately upon learning of the event.

Serious Adverse Event (SAE) – An SAE is any adverse event that led to any of the following:

- Death
- Serious deterioration in the health of the subject that resulted in any of the following:
- Life-threatening illness or injury
- Permanent or persistent impairment of a body structure or a body function
- Hospitalization or prolongation of patient hospitalization
- Medical or surgical intervention to prevent life-threatening illness or injury or permanent impairment to a body structure or a body function.
- Chronic disease
- Fetal distress, fetal death or a congenital physical or mental impairment of birth defect.

Diagnoses and conditions that are considered Ocular Serious Adverse Events include, but not limited to:

- Microbial Keratitis (MK)
- Iritis (including cells in the anterior chamber)
- Permanent decrease in best spectacle corrected visual acuity equivalent to 2 acuity lines or greater
- Central Corneal Opacity
- Central Corneal Neovascularization
- Uveitis
- Endophthalmitis
- Hypopyon
- Hyphemia
- Penetration of Bowman's Membrane
- Persistent Epithelial Defect
- Limbal cell Damage leading to Conjunctivalization

**Significant Adverse Events** – are defined as events that are symptomatic and warrant discontinuation (temporary or permanent) of the contact lens wear

Diagnoses and conditions that are considered Ocular Significant Adverse Events include, but not limited to the following:

- Contact Lens Induced Peripheral Ulcer (CLPU)
- Significant Infiltrative Events (SIE)
- Superior Epithelial Arcuate Lesions (SEALs)
- Any Temporary Loss of > 2 Lines of BSCVA
- Other grade 3 or higher corneal findings, such as abrasions or edema
- Non-contact lens related corneal events e.g. Epidemic Keratoconjunctivitis (EKC)
- Asymptomatic Corneal Scar
- Any corneal event which necessitates temporary lens discontinuation > 2 weeks

**Non-Significant Adverse Events** – are defined as those events that are usually asymptomatic and usually do not warrant discontinuation of contact lens wear but may cause a reduction in wear time. However, the Investigator may choose to prescribe treatment as a precautionary measure.

Diagnoses and conditions that are considered Ocular Non-Significant Adverse Events include, but not limited to the following:

- Non-significant Infiltrative Event (NSIE)
- Contact Lens Papillary Conjunctivitis (CLPC)
- Superficial Punctate Keratitis (SPK)
- Conjunctivitis: Bacterial, Viral, Allergic
- Blepharitis
- Meibomianitis
- Contact Dermatitis

- Localized Allergic Reactions
- Any corneal event not explicitly defined as serious or significant adverse event, which necessitates temporary lens discontinuation < 2 weeks

**Adverse Device Effect (ADE)** – An ADE is an "adverse event related to the use of an investigational medical device.

**NOTE 1:** to entry: This definition includes adverse events resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational medical device.

NOTE 2 to entry: This definition includes any event resulting from use error or from intentional misuse of the investigational medical device."

Unanticipated Adverse Device Effect (UADE) – Any serious adverse effect on health or safety or any life-threatening problem or death caused by, or associated with, the test article, if that effect, problem, or death was not previously identified in nature, severity, or degree of incidence in the investigational plan, Investigator's Brochure or protocol, or any other unanticipated serious problem associated with the test article that relates to the rights, safety and welfare of subjects.

#### 13.2. Assessing Adverse Events

In conjunction with the medical monitor, the Investigator will evaluate adverse events to ensure the events are categorized correctly. Elements of categorization will include:

- Seriousness/Classifications (see definition in Section 13.1).
- Causality or Relatedness i.e. the relationship between the test article, study treatment or study procedures and the adverse event (not related; unlikely related; possibly related; related see definition in Section 13.2.1).
- Adverse Event Severity Adverse event severity is used to assess the degree of intensity of the adverse event (mild; moderate; severe for all events see definition in Section 13.2.2).
- Outcome not recovered or not resolved; recovering or resolving; recovered or resolved with sequelae; recovered or resolved; death related to adverse event; unknown.
- Actions Taken none; temporarily discontinued; permanently discontinued; other.

#### 13.2.1. Causality Assessment

**Causality Assessment** – A determination of the relationship between an adverse event and the test article. The test article relationship for each adverse event should be determined by the investigator using these explanations:

- Not Related- An adverse event that is not related to the use of the test article, study treatment or study procedures.
- Unlikely Related An adverse event for which an alternative explanation is more likely, e.g. concomitant treatment, concomitant disease(s), or the relationship of time suggests that a causal relationship is not likely.

- Possibly Related An adverse event that might be due to the use of the test article, or to the study treatment or study procedures. An alternative explanation, e.g. concomitant treatment, concomitant disease(s), is inconclusive. The relationship in time is reasonable. Therefore, the causal relationship cannot be excluded.
- Related An adverse event that is listed as a possible adverse effect (device) or adverse reaction (drug) and cannot be reasonably explained by an alternative explanation, e.g. concomitant treatment of concomitant disease(s). The relationship in time is very suggestive, e.g. it is confirmed by de-challenge and re-challenge.

#### 13.2.2. Severity Assessment

**Severity Assessment** – A qualitative assessment of the degree of intensity of an adverse event as determined by the Investigator or reported to him/her by the subject. The assessment of severity is made irrespective of test article, study treatment or study procedure relationship or seriousness of the event and should be evaluated according to the following scale:

- Mild Event is noticeable to the subject, but is easily tolerated and does not interfere with the subject's daily activities.
- Moderate Event is bothersome, possible requiring additional therapy, and may interfere with the subject's daily activities.
- Severe Event is intolerable, necessitates additional therapy or alteration of therapy and interferes with the subject's daily activities.

#### 13.3. Documentation and Follow-Up of Adverse Events

The recording and documenting of adverse events (ocular and non-ocular) begin when the subjects are exposed to the test article, study treatment or study procedure. Adverse events reported before the use of test article, start of study treatment, or study procedures will be recorded as medical history. However, if the condition deteriorates at any time during the study it will be recorded and reported as an AE. Untoward medical events reported after the subject's exit from the study will be recorded as adverse events at the discretion of the Investigator.

Upon finding an adverse event, the Principal Investigator will document the condition in the subject record and in the eCRFs. He/she will complete the Adverse Event /eCRF.

Complete descriptions of all adverse events must be available in the subject record. All Adverse Events including local and systemic reactions not meeting the criteria for "serious adverse events" shall be captured on the appropriate case report form or electronic data system. All adverse events occurring while the subject is enrolled in the study must be documented appropriately regardless of relationship.

It is the Investigator's responsibility to maintain documentation of each reported adverse event. All adverse events will be followed in accordance with applicable licensing requirements. Such documentation will include the following:

- Adverse event (diagnosis not symptom).
- Drawings or photographs (where appropriate) that detail the finding (e.g., size, location, and depth, etc.).
- Date the clinical site was notified.
- Date and time of onset.
- Date and time of resolution.
- Adverse event classification, severity, and relationship to test articles, as applicable.
- Treatment regimen instituted, including concomitant medications prescribed, in accordance with applicable licensing requirements.
- Any referral to another health care provider if needed.
- Outcome, ocular damage (if any).
- Likely etiology.
- Best corrected visual acuity at the discovery of the event and upon conclusion of the event.

In addition, if an infiltrate(s) is present, he/she will complete the Corneal Infiltrate Assessment eCRF. Where necessary, a culture of the corneal lesion will be collected to determine if the infection is microbial in nature. If cultures are collected, the date of culture collection and laboratory utilized will be recorded.

Changes in the severity of an AE shall be documented to allow an assessment of the duration of the event at each level of intensity to be performed. Adverse events characterized as intermittent require documentation of the onset and duration of each episode. Changes in the assessment of relationship to the Test Article shall also be clearly documented.

Subjects who present with an adverse event shall be followed by the Investigator, within licensure, until all signs and symptoms have returned to pre-treatment status, stabilized, or been satisfactorily resolved. If further treatment beyond licensure is required, the patient will be referred to the appropriate health care provider. The Investigator will use his/her clinical judgment as to whether a subject reporting with an adverse event will continue in the study. If a subject is discontinued from the study, it will be the responsibility of the Investigator to record the reason for discontinuation. The Investigator will also document the adverse event appropriately and complete the Adverse Event eCRF. Any subjects with ongoing adverse events related to the test article, study treatment or study procedures, as of the final study visit date, should be followed to resolution of the adverse event or until referral to an appropriate health care provider, as recommended by the Investigator. Non-ocular adverse events that are not related to the test article, study treatment, or study procedures may be recorded as "ongoing" without further follow-up.

#### 13.4. Reporting Adverse Events

The Investigator will notify the Sponsor of an adverse event by e-mail, facsimile, or telephone as soon as possible and no later than 24 hours from discovery for any serious /significant adverse events, and 2 days from discovery for any non-significant adverse event. In addition, a written report will be submitted by the Principal Investigator to the IEC/IRB according to their requirements (Section 13.4.2). The report will comment whether the adverse event was considered to be related to the test article, study treatment or study procedures.


# 13.4.1. Reporting Adverse Events to Sponsor

#### Serious/Significant Adverse Events

The Investigator will inform the sponsor of all serious/significant adverse events occurring during the study period as soon as possible by e-mail, fax, or telephone, but no later than 24 hours following discovery of the event. The Investigator is obligated to pursue and obtain information requested by the Sponsor in addition to that information reported on the eCRF. All subjects experiencing a serious/significant adverse event must be followed up and all outcomes must be reported.

When medically necessary, the Investigator may break the randomization code to determine the identity of the treatment that the subject received. The Sponsor and study monitor should be notified prior to unmasking the test articles.

In the event of a serious/significant adverse event, the Investigator must:

- Notify the Sponsor immediately.
- Obtain and maintain in the subject's records all pertinent medical information and medical judgment for colleagues who assisted in the treatment and follow-up of the subject.
- Provide the Sponsor with a complete case history which includes a statement as to whether the event was or was not related to the use of the test article.
- Notify the IEC/IRB as required by the IEC/IRB reporting procedure according to national regulations.

#### **Unanticipated (Serious) Adverse Device Effect (UADE)**

In the event of an Unanticipated (Serious) Adverse Device Effect (UADE), the Investigator will submit a report of the UADE to the Sponsor and IEC/IRB as soon as possible, but no later than 24 hours after the Investigator first learns of the effect. This report is in addition to the immediate notification mentioned above.

The Sponsor must conduct an evaluation of the UADE and must report the results of the evaluation to FDA, the IEC/IRB and participating Investigators within 10 working days after the Sponsor first receives notification of the effect.

#### **Non-Serious Adverse Events**

All non-serious adverse events, including non-serious adverse device effects, will be reported to the sponsor by the Investigator no later than 2 days from discovery.

#### 13.4.2. Reporting Adverse Events to the Responsible IEC/IRB and Health Authorities

Adverse events that meet the IEC/IRB requirements for reporting must be reported within the IEC/IRB's written guidelines. Each clinical site will refer to and follow any guidelines set forth by their Approving IEC/IRB. Each clinical site will refer to and follow any guidelines set forth by their local governing Health Authorities.

The Sponsor will report applicable Adverse Events to the local health authorities according the written guidelines, including reporting timelines.

#### 13.4.3. Event of Special Interest

None

#### 13.5. Reporting of Pregnancy

Subjects reporting pregnancy (by self-report) during the study will be discontinued after the event is recorded as an Adverse Event. Once discontinued, pregnant participants and their fetuses will not be monitored for study related purposes.

Pregnant participants are not discontinued from contact lens or solution related studies for safety concerns, but due to general concerns relating to pregnancy and contact lens use. Specifically, pregnant women are discontinued due to fluctuations in refractive error and/or visual acuity that occur secondary to systemic hormonal changes, and not due to unforeseen health risks to the mother or fetus.

#### 14. STATISTICAL METHODS

#### 14.1. General Considerations

Statistical Analysis will be undertaken by the sponsor or under the authority of the sponsor. A general description of the statistical methods to be implemented in this clinical trial is outlined below.

All data summaries and statistical analyses will be performed using the SAS software Version 9.4 or higher (SAS Institute, Cary, NC)<sup>7</sup>. Throughout the analysis of data, the results for each subject/eye will be used when available for summarization. Unscheduled visits will be summarized separately.

Summary tables (descriptive statistics and/or frequency tables) will be provided for all baseline variables, efficacy variables and safety variables as appropriate. Continuous variables will be summarized with descriptive statistics (n, mean, standard deviation [SD]), median, minimum and maximum). Frequency count and percentage of subjects or eyes within each category will be provided for categorical data.

#### 14.2. Sample Size Justification

Approximately 30 subjects will be enrolled in this study to attain a minimum of 25 completed subjects. This is a feasibility descriptive study to evaluate the visual acuity after the instillation of a lipid-based eye drop. Sample size is not based on the empirical power analysis, and the data collected for this study may be used in future study design if applicable.

#### 14.3. Analysis Populations

#### **Safety Population:**

All subjects who were administered any test article excluding subjects who drop out prior to administering any test article. At least one observation should be recorded.

#### **Per-Protocol Population:**

All subjects who have successfully completed all visits and did not substantially deviate from the protocol as determined by the trial cohort review committee prior to database hard lock. Justification of excluding subjects with protocol deviations in the Per-Protocol Population set will be documented in a memo to file.

#### **Intent-to-Treat (ITT) Population:**

All randomized subjects regardless of actual treatment and subsequent withdrawal from study or deviation from protocol. At least one observation should be recorded.

#### 14.4. Level of Statistical Significance

No inferential statistics are planned to be performed in this study; hence, the level of statistical significance is not a concern. In the event that exploratory analysis is conducted, an overall type I error rate of 5% will be used.

#### 14.5. Primary Analysis

Change in logMAR visual acuity will be descriptively summarized.

#### 14.6. Secondary Analysis

Not applicable.

#### 14.7. Other Exploratory Analyses

The following study endpoints will be disruptively summarized:

- Slit Lamp Findings using FDA scale
- Snellen best corrected distance visual acuity
- Subject reported ocular symptoms
- Adverse Events
- Number and reasons for discontinuation will be monitored.

#### 14.8. Interim Analysis

Not applicable.

#### 14.9. Procedure for Handling Missing Data and Drop-Outs

Missing or spurious values will not be imputed. The count of observed values will be included in the summary tables and listings.

#### 14.10. Procedure for Reporting Deviations from Statistical Plan

The analysis will be conducted according to that specified in above sections. There are no known reasons for which it is planned to deviate from these analysis methods. If for any reason a change is made, the change will be documented in the study report along with a justification for the change.

#### 15. DATA HANDLING AND RECORD KEEPING/ARCHIVING

#### 15.1. Electronic Case Report Form/Data Collection

The data for this study will be captured on electronic case report forms (eCRFs) using an EDC system (Bioclinica 5.5). An authorized data originator will enter study data into the eCRFs using the EDC system. Data collected on equipment that is not captured in EDC will be formatted to the specification of the JJVC database manager and sent to JJVC for analysis.

External Data Sources for this study include: Not applicable.

The clinical data will be recorded on dedicated eCRFs specifically designed to match the study procedures for each visit. Only specifically delegated staff can enter data on a CRF. Once completed, the eCRFs will be reviewed for accuracy and completeness and signed by the Investigator. The sponsor or sponsor's representatives will be authorized to gain access to the subject recordation for the purposes of monitoring and auditing the study.

Edit checks, electronic queries, and audit trails are built into the system to ensure accurate and complete data collection. Data will be transmitted from the clinical site to a secure central database as forms are completed or updated, ensuring information accuracy, security, and confidentiality. After the final database lock, the Investigator will be provided with Individual Patient Profiles (IPP) including the full audit trail on electronic media in PDF format for all of the study data. The IPP must be retained in the study files as a certified copy of the source data for the study.

The content and structure of the eCRFs are compliant with ISO14155:2011.<sup>1</sup>

#### 15.2. Subject Record

At a minimum, subject record should be available for the following:

- subject identification
- eligibility
- study identification
- study discussion
- provision of and date of informed consent
- visit dates
- results of safety and efficacy parameters as required by the protocol
- a record of all adverse events
- follow-up of adverse events
- medical history and concomitant medication
- test article receipt/dispensing/return records
- date of study completion
- reason for early discontinuation of test article or withdrawal from the study, if applicable

The subject record is the eCRF or an external record. The author of an entry in the subject record must be identifiable. The first point of entry is considered to be the source record.

Adverse event notes must be reviewed and initialed by the Investigator.

#### 15.3 ClinicalTrials.gov

This pilot study is being conducted after final formulation and meets the criteria for registration.

#### 16. DATA MANAGEMENT

#### 16.1. Access to Source Data/Document

The Investigator/Institution will permit trial-related monitoring, audits, IEC/IRB review and regulatory inspection(s) by providing direct access to source data/documents. Should the clinical site be contacted for an audit by an IEC/IRB or regulatory authority, JJVC must be contacted and notified in writing within 24 hours.

#### 16.2. Confidentiality of Information

Information concerning the investigational product and patent application processes, scientific data or other pertinent information is confidential and remains the property of JJVC. The Investigator may use this information for the purposes of the study only. It is understood by the Investigator that JJVC will use information developed in this clinical study in connection with the development of the investigational product and therefore may disclose it as required to other clinical investigators and to regulatory agencies. In order to allow the use of the information derived from this clinical study, the Investigator understands that he/she has an obligation to provide complete test results and all data developed during this study to the Sponsor.

#### 16.3. Data Quality Assurance

Steps will be taken to ensure the accuracy and reliability of data, include the selection of qualified investigators and appropriate clinical sites and review of protocol procedures with the Principal Investigator. The Principal Investigator, in turn, must ensure that all Sub-Investigators and clinical site personnel are familiar with the protocol and all study-specific procedures and have appropriate knowledge of the study article.

Training on case report form completion will be provided to clinical site personnel before the start of the study. The Sponsor will review case report forms for accuracy and completeness remotely during the conduct of the study, during monitoring visits, and after transmission to data management. Any data discrepancies will be resolved with the Investigator or designee, as appropriate.

Quality Assurance representatives from JJVC may visit clinical sites to review data produced during the study and to access compliance with applicable regulations pertaining to the conduct

of clinical trials. The clinical sites will provide direct access to study-related source data/documents and reports for the purpose of monitoring and auditing by JJVC and for inspection by local and regulatory authorities.

#### 17. CLINICAL MONITORING

The study monitors will maintain close contact with the Principal Investigator and the Investigator's designated clinical site personnel. The monitor's responsibilities will include:

- Ensuring that the investigation is being conducted according to the protocol, any subsequent versions, and regulatory requirements are maintained.
- Ensuring the rights and wellbeing of subjects are protected.
- Ensuring adequate resources, including facilities, laboratories, equipment, and qualified clinical site personnel.
- Ensuring that protocol deviations are documented with corrective action plans, as applicable.
- Ensuring that the clinical site has sufficient test article and supplies.
- Clarifying questions regarding the study.
- Resolving study issues or problems that may arise.
- Reviewing of study records and source documentation verification in accordance with the monitoring plan.

#### 18. ETHICAL AND REGULATORY ASPECTS

#### 18.1. Study-Specific Design Considerations

Potential subjects will be fully informed of the risks and requirements of the study and, during the study, subjects will be given any new information that may affect their decision to continue participation. Subjects will be told that their consent to participate in the study is voluntary and may be withdrawn at any time with no reason given and without penalty or loss of benefits to which they would otherwise be entitled. Only subjects who are fully able to understand the risks, benefits, and potential adverse events of the study, and provide their consent voluntarily will be enrolled.

#### 18.2. Investigator Responsibility

The Principal Investigator is responsible for ensuring that the clinical study is performed in accordance with the signed agreement, the investigational plan, Section 4 of the ICH E6 guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements. GCP is an international ethical and scientific quality standard for designing, conducting, recording, and reporting studies that involve the participation of human subjects. Compliance with this standard provides public assurance that the rights, safety, and well-being of study subjects are protected, consistent with the principles of the Declaration of Helsinki 64<sup>th</sup> WMA General Assembly 2013<sup>3</sup> and that the clinical study data are credible. The Investigator must maintain clinical study files in accordance with Section 8 of the ICH E6 guidelines on Good Clinical Practice (GCP),<sup>2</sup> and applicable regulatory requirements.

#### 18.3. Independent Ethics Committee or Institutional Review Board (IEC/IRB)

Before the start of the study, the Investigator (or Sponsor when applicable) will provide the IEC/IRB with current and complete copies of the following documents (where applicable):

- Final protocol.
- Sponsor-approved informed consent form (and any other written materials to be provided to the subjects)
- Investigator's Brochure (or equivalent information).
- Sponsor-approved subject recruitment materials.
- Information on compensation for study-related injuries or payment to subjects for participation in the study.
- Investigator's curriculum vitae, clinical licenses, or equivalent information (unless not required, as documented by IEC/IRB).
- Information regarding funding, name of the Sponsor, institutional affiliations, other potential conflicts of interest, and incentives for subjects.
- Any other documents that the IEC/IRB requests to fulfill its obligation.

This study will be undertaken only after IEC/IRB has given full approval of the final protocol, the informed consent form, applicable recruiting materials, and subject compensation programs, and the Sponsor has received a copy of this approval. This approval letter must be dated and must clearly identify the documents being approved.

During the study, the Investigator (or Sponsor when applicable) will send the following documents to the IEC/IRB for their review and approval, where appropriate:

- Protocol revisions
- Revision(s) to informed consent form and any other written materials to be provided to subjects
- If applicable, new or revised subject recruitment materials approved by the Sponsor
- Revisions to compensation for study-related injuries or payment to subjects for participation in the study
- Investigator's Brochure revisions
- Summaries of the status of the study (at least annually or at intervals stipulated in guidelines of the IEC/IRB)
- Reports of adverse events that are serious, unanticipated, and associated with the test articles, according to the IRB's requirements
- New information that may adversely affect the safety of the subjects or the conduct of the study
- Major protocol deviations as required by the IEC/IRB
- Report of deaths of subjects under the Investigator's care
- Notification if a new Investigator is responsible for the study at the clinical site
- Any other requirements of the IEC/IRB

For protocol revisions that increase subject risk, the revisions and applicable informed consent form revisions must be submitted promptly to the IEC/IRB for review and approval before implementation of the change(s).

At least once a year, the IEC/IRB will review and reapprove this clinical study. This request should be documented in writing.

At the end of the study, the Investigator (or Sponsor where required) will notify the IEC/IRB about the study completion. Documentation of this notification must be retained at the clinical site and a copy provided to the CRO or Sponsor as applicable.

#### 18.4. Informed Consent

Each subject or their representative, must give written consent according to local requirements after the nature of the study has been fully explained. The consent form must be signed before performance of any study-related activity. The consent form that is used must be approved by both the Sponsor and by the reviewing IEC/IRB. The informed consent is in accordance with principles that originated in the Declaration of Helsinki,<sup>3</sup> current ICH<sup>2</sup> and ISO 14155<sup>1</sup> guidelines, applicable regulatory requirements, and Sponsor Policy.

Before entry into the study, the Investigator or an authorized member of the clinical site personnel must explain to potential subject the aims, methods, reasonably anticipated benefits, and potential hazards of the study, and any discomfort it may entail. Subjects will be informed that their participation is voluntary and that they may withdraw consent to participate at any time.

The subject will be given sufficient time to read the informed consent form and the opportunity to ask questions. After this explanation and before entry into the study, consent should be appropriately recorded by means of the subject's dated signature. After having obtained the consent, a copy of the informed consent form must be given to the subject.

#### 18.5. Privacy of Personal Data

The collection, processing and disclosure of personal data and medical information related to the Study Subject, and personal data related to Principal Investigator and any clinical site personnel (e.g., name, clinic address and phone number, curriculum vitae) is subject to compliance with the Health Information Portability and Accountability Act (HIPAA) in the United States<sup>5</sup> and other applicable personal data protection and security laws and regulations. Appropriate measures will be employed to safeguard these data, to maintain the confidentiality of the person's related health and medical information, to properly inform the concerned persons about the collection and processing of their personal data, to grant them reasonable access to their personal data and to prevent access by unauthorized persons.

All information obtained during the course of the investigation will be regarded as confidential. All personal data gathered in this trial will be treated in strictest confidence by Investigators, monitors, Sponsor's personnel and IEC/IRB. No data will be disclosed to any third party without the express permission of the subject concerned, with the exception of Sponsor personnel (monitor, auditor), IEC/IRB and regulatory organizations in the context of their

investigation related activities that, as part of the investigation will have access to the CRFs and subject records.

The collection and processing of personal data from subjects enrolled in this study will be limited to those data that are necessary to investigate the efficacy, safety, quality, and utility of the investigational product(s) used in this study.

These data must be collected and processed with adequate precautions to ensure confidentiality and compliance with applicable data privacy protection laws and regulations.

The Sponsor ensures that the personal data will be:

- processed fairly and lawfully.
- collected for specified, explicit, and legitimate purposes and not further processed in a way incompatible with these purposes.
- adequate, relevant, and not excessive in relation to said purposes.
- accurate and, where necessary, kept current.

Explicit consent for the processing of personal data will be obtained from the participating subject before collection of data. Such consent should also address the transfer of the data to other entities and to other countries.

The subject has the right to request through the Investigator access to his personal data and the right to request rectification of any data that are not correct or complete. Reasonable steps should be taken to respond to such a request, taking into consideration the nature of the request, the conditions of the study, and the applicable laws and regulations.

Appropriate technical and organizational measures to protect the personal data against unauthorized disclosures or access, accidental or unlawful destruction, or accidental loss or alteration must be put in place. Sponsor personnel whose responsibilities require access to personal data agree to keep the identity of study subjects confidential.

#### 19. STUDY RECORD RETENTION

In compliance with the ICH/GCP guidelines,<sup>2</sup> the Investigator/Institution will maintain all CRFs and all subject records that support the data collected from each subject, as well as all study documents as specified in ICH/GCP<sup>2</sup> and all study documents as specified by the applicable regulatory requirement(s). The Investigator/Institution will take measures to prevent accidental or premature destruction of these documents.

Essential documents must be retained until at least two (2) years after the last approval of a marketing application in an ICH region and until there are no pending or contemplated marketing applications in an ICH region or until at least two (2) years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents will be retained for a longer period if required by the applicable regulatory requirements or instructed by the Sponsor. It is the responsibility of the Sponsor to inform the Investigator/Institution as to when these documents no longer need to be retained.

If the responsible Investigator retires, relocates, or for other reasons withdraws from the responsibility of keeping the study records, custody must be transferred to a person who will accept the responsibility. The Sponsor must be notified in writing of the name and address of the new custodian. Under no circumstance shall the Investigator relocate or dispose of any study documents before having obtained written approval from the Sponsor.

If it becomes necessary for the Sponsor or the appropriate regulatory authority to review any documentation relating to this study, the Investigator must permit access to such reports. If the Investigator has a question regarding retention of study records, he/she should contact JJVC.

#### 20. FINANCIAL CONSIDERATIONS

Remuneration for study services and expenses will be set forth in detail in the Clinical Research Agreement. The Research Agreement will be signed by the Principal Investigator and a JJVC management representative prior to study initiation.

JJVC reserves the right to withhold remuneration for costs associated with protocol violations such as:

- Continuing an ineligible subject in the study.
- Scheduling a study visit outside the subject's acceptable visit range.

JJVC reserves the right to withhold final remuneration until all study related activities have been completed, such as:

- Query resolution.
- Case Report Form signature.
- Completion of any follow-up action items.

#### 21. PUBLICATION

This study will be registered on ClinicalTrials.gov based on the following: this study is being conducted after final formulation lock.

#### 22. REFERENCES

- 1. ISO 14155:2011: Clinical Investigation of Medical Devices for Human Subjects Good Clinical Practice. Available at: https://www.iso.org/standard/45557.html
- 2. International Conference on Harmonization Good Clinical Practice E6 (ICH-GCP). Available at: http://www.ich.org/products/guidelines/efficacy/article/efficacy-guidelines.html
- 3. Declaration of Helsinki Ethical principles for Medical Research Involving Human Subjects. Available at: https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects/
- 4. United States (US) Code of Federal Regulations (CFR). Available at: https://www.gpo.gov/fdsys/browse/collectionCfr.action?collectionCode=CFR
- 5. Health Information Portability and Accountability Act (HIPAA). Available at: https://www.hhs.gov/hipaa/for-professionals/privacy/index.html
- 6. EU MDR 2017/745
- 7. SAS Institute Inc. 2016 SAS/STAT® 14.3 User's Guide. Cary, NC: SAS Institute Inc.

# **APPENDIX A: PATIENT INSTRUCTION GUIDE**

A Clinic Only Wear Patient Instruction Guide will be provided separately.

APPENDIX B: PACKAGE INSERT (APPROVED PRODUCT)



**Lubricating Eye Drops** 

# **Drug Facts**

# **Active Ingredient**

**Purpose** 

Polyethylene Glycol 400 0.25% . . . . . Eye lubricant

**Uses** ■ For the temporary relief of burning, irritation, and discomfort due to dryness of the eye or exposure to wind or sun.

■ May be used as a protectant against further irritation.

# **Warnings**

- For external use only.
- To avoid contamination, do not touch tip of container to any surface. Replace cap after using.
- Do not use if solution changes color or becomes cloudy.

#### Stop use and ask a doctor if:

You experience eye pain, changes in vision, continued redness or irritation of the eye, or if the condition worsens or persists for more than 72 hours.

# Keep out of the reach of children.

If swallowed, get medical help or contact a Poison Control Center right away.

#### **Directions**

Instill 1 or 2 drops in the affected eye(s) as needed or as directed by your eye care professional.

# *Inactive Ingredients*

Boric Acid; Calcium Chloride; Magnesium Chloride; Potassium Chloride; Purified Water; Sodium Borate; Sodium Chloride; Sodium Chlorite (OcuPure® brand) as a preservative; Sodium Hyaluronate.

# Other Information

Use only if tape seals on top and bottom flaps are intact. RETAIN THIS CARTON FOR FUTURE REFERENCE.

Discard solution 90 days after opening

Product of China made in accordance with US FDA guidelines Blink is a trademark of Johnson & Johnson Surgical Vision, Inc.

© Johnson & Johnson Surgical Vision, Inc. 2017 Santa Ana, CA 92705

No. 93286BT

AM60870US12C 9587X

Revision Date: 07/2018

JJVC CONFIDENTIAL CR-6371, v4.0 Page 51 of 86

# APPENDIX C: SUBJECT REPORTED OCULAR SYMPTOMS BIOMICROSCOPY SCALE DISTANCE AND NEAR VISUAL ACUITY EVALUATION ETDRS DISTANCE VISUAL ACUITY MEASURMENT PROCEDURE VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINATION TESTING

SUBJECT REPORTED OCULAR SYMPTOMS

Subject Reported Ocular Symptoms/Problems Title: Document Type: Document Number: Revision Number: 3



# Johnson & Johnson Vision Care, Inc.


DISTANCE AND NEAR VISUAL ACUITY EVALUATION

Johnson & Johnson Vision Care, Inc. Distance and Near Snellen Visual Acuity Evaluation Title: Document Type: Document Number: **Revision Number: 4** 

Johnson & Johnson Vision Care, Inc. Distance and Near Snellen Visual Acuity Evaluation Title: **Document Type: Document Number: Revision Number: 4** 

Johnson & Johnson Vision Care Inc Distance and Near Snellen Visual Acuity Evaluation Title: **Document Type:** Document Number: **Revision Number: 4** 

JJVC CONFIDENTIAL

Title: Distance and Near Snellen Vision Care, Inc.
Document Type: Revision Number: 4



ETDRS DISTANCE VISUAL ACUITY MEASUREMENT PROCEDURE

# Johnson & Johnson Vision Care, Inc.

Distance LogMAR Visual Acuity Measurement Procedure Title: Document Type: **Document Number: Revision Number: 4** 

# Johnson & Johnson Vision Care, Inc.

| Title: | Distance LogMAR Visual Acuity Measurement Procedure | |
|---|---|---|
| Document Type: | | - 20 |
| Document Number: | | Revision Number: 4 |



# Johnson & Johnson Vision Care, Inc.



VISUAL ACUITY CHART LUMINANCE AND ROOM ILLUMINATION

# Johnson & Johnson Vision Care, Inc.

Visual Acuity Chart Luminance and Room Illumination Testing Title: **Document Type: Document Number:** Revision Number: 3

# Johnson & Johnson Vision Care, Inc.

Title: Visual Acuity Chart Luminance and Room Illumination Testing

Document Type: Revision Number: 3


## **Clinical Study Protocol**

## Johnson & Johnson Vision Care, Inc.

| Title: | Visual Aculty Chart Luminance and Room Humination Testing |
|------------------|-----------------------------------------------------------|
| Document Type: | |
| Document Number: | Revision Number: 3 |

### **Clinical Study Protocol**

### Johnson & Johnson Vision Care, Inc.

Visual Acuity Chart Luminance and Room Illumination Testing Title: **Document Type:** Document Number: **Revision Number: 3** 

## **Clinical Study Protocol**

### Johnson & Johnson Vision Care, Inc.

| Title: | Visual Acuity Chart Luminance | and Room Illumination Testing |
|---|---|---|
| Document Type: | | |
| Document Number: | * | Revision Number: 3 |
| | | <del></del> |
| 4 | | |
| | i i | |

APPENDIX D: GUIDELINES FOR COVID-19 RISK MITIGATION

# Clinical Study Protocol Johnson & Johnson Vision Care, Inc. Guidelines for COVID 19 Risk Mitigation

| Title: | Guidennes for COVID-19 Risk Mingation | JV1D-19 RISK MILIGATION |
|---|---|---|
| Document Type: | and a | |
| Document Number | | Revision Number 1 |

#### 1.0 PURPOSE

The purpose of this document is to provide guidelines for the re-opening or initiation of clinical study sites in the United States (US) participating in Johnson & Johnson Vision Care, Inc. (JJVCI) clinical studies during the COVID-19 pandemic.

#### 2.0 SCOPE

This document provides guidelines for Johnson & Johnson Vision Care (JJVCI) to address the potential risks from COVID-19 to study subjects, investigators, study site staff, and monitors at study sites in the US. These guidelines do not apply to study sites outside of the US. The guidance provided in this document is in effect from the date of approval through the date of retirement of this Work Instruction. At a minimum, this Work Instruction will be reviewed and updated on a quarterly basis, as appropriate.

NOTE: Sites outside of the US will be evaluated on a site by site basis subject to local health authority guidance.

#### 3.0 DEFINITIONS

American Academy of Optometry (AAO): The American Academy of Optometry is an organization of optometrists based in Orlando, Florida. Its goal is to maintain and enhance excellence in optometric practice, by both promoting research and the dissemination of knowledge. The AAO holds an annual meeting, publishes a monthly scientific journal, gives credentials to optometrists through the fellowship process and publishes position statements.

American Optometric Association (AOA): The American Optometric Association, founded in 1898, is the leading authority on quality care and an advocate for our nation's health, representing more than 44,000 doctors of optometry (O.D.), optometric professionals, and optometry students. Doctors of optometry take a leading role in patient care with respect to eye and vision care, as well as general health and well-being. As primary health care providers, doctors of optometry have extensive, ongoing training to examine, diagnose, treat and manage ocular disorders, diseases and injuries and systemic diseases that manifest in the eye. The American Optometric Association is a federation of state, student, and armed forces optometric associations. Through these affiliations, the AOA serves members consisting of optometrists, students of optometry, paraoptometric assistants and technicians. The AOA and its affiliates work to provide the public with quality vision and eye care.

Center for Disease Control (CDC): The Centers for Disease Control and Prevention is a national public health institute in the United States. It is a United States federal agency, under the Department of Health and Human Services, and is headquartered in Atlanta, Georgia.

**COVID-19:** Current outbreak of respiratory disease caused by a novel coronavirus. The virus has been named "SARS-CoV-2" and the disease it causes has been named "Coronavirus Disease 2019" (COVID-19).

Clinical Study: Voluntary research studies conducted in people and designed to answer specific questions about the safety or effectiveness of drugs, vaccines, other therapies, or new ways of using existing treatments. May also be called clinical trials, studies, research, trials, or protocols.

Clinical Study Site: Location where a clinical study is conducted, such as a doctor's office, university, or laboratory. Clinical studies are conducted by Investigators who are individual(s) responsible for the conduct of the clinical study at a study site. If a study is conducted by a team of individuals, the Investigator is the responsible leader of the team and may be called the Principal Investigator.

Clinical Operations Manager (COM): The Johnson & Johnson Vision Care (JJVCI) individual responsible for the overall management of a clinical trial.


## Clinical Study Protocol Johnson & Johnson Vision Care, Inc. Chidelines for COVID 10 Pick Mitigation

Title: Guidelines for COVID-19 Risk Mitigation

Document Type: Revision Number: 1

**Monitor:** An individual designated to oversee the progress of a clinical study and ensure that it is conducted, recorded, and reported in accordance with the protocol, Standard Operating Procedures (SOPs), Good Clinical Practice (GCP), and applicable regulatory requirements.

Medical Safety Officer (MSO): Physician who has primary accountability in their product portfolio for product health and safety, and who serves as an independent medical voice for patient safety.

**Safety Management Team (SMT):** A cross-functional, collaborative team responsible for review, assessment and evaluation of medical safety data arising from any source throughout the product life cycle.

#### 4.0 GUIDANCE FOR STUDY DOCUMENTS

In alignment with recent health authority guidance, JJVCI is providing recommendations for study-related management in the event of disruption to the conduct of the clinical study. This guidance does not supersede any local or government requirements or the clinical judgement of the investigator to protect the health, safety and well-being of participants and site staff. If, at any time, a participant's safety is considered to be at risk, study intervention will be discontinued, and study follow-up will be conducted as outlined in the protocol.

During the COVID-19 pandemic, the additional risks listed below need to be considered for study participants and study personnel:

#### 4.1 Additional Risks Related to the COVID-19 Pandemic:

- The possible transmission of the Coronavirus infection and consequent complications, beyond the risk of adverse events due to the investigational device and/or procedures.
- The risk may be higher in an optometric clinical study because of the close contact the subject will have with health care professionals during the procedures and assessments (since the investigator must make the measurements close to the subject's face) and, in addition the need for multiple follow-up visits/exams which may expose the subject to other patients and/or healthcare professionals who might be transmitting the virus, even if they do not have symptoms.
- Potential disruptions to the study may be necessary due to current or future pandemic-related emergency restrictions, which may lead to delays in scheduled follow-up visits.
- Subjects experiencing an adverse event related to contact lens wear may receive delayed treatment
  due to COVID-19 restrictions. In this event, all assessments that can be conducted virtually will be
  completed by the investigator to determine the best course of treatment for the subject, including
  an unscheduled visit, up to discontinuation from the study, as appropriate.

If a study subject is found to have contracted COVID-19 during participation in a study, he/she will be discontinued from the study and followed until COVID-19 Adverse Event (AE) resolution.

To help minimize the above potential risks, JJVCI recommend reviewing/complying with local, state, and governmental guidance for COVID-19 risks.

JJVCI will provide the following study specific documents with language pertaining to COVID-19 risks:

#### 4.1.1 Informed Consent:

Will include information concerning the study-associated risks related to the COVID-19 pandemic in bold font and/or boxed on the first page of the Informed Consent document:


## Clinical Study Protocol Johnson & Johnson Vision Care, Inc. Cuidelines for COVID 10 Pick Mitigation

Title: Guidelines for COVID-19 Risk Mitigation

Document Type: Revision Number: 1

#### STUDY ASSOCIATED RISKS RELATED TO COVID-19 (CORONAVIRUS) PANDEMIC

It is important to note that this study will be conducted, at least in part, during the COVID-19 pandemic. As such, additional risks associated with the infection with COVID-19 exist for you. This is particularly important for this study due, in part, to the closeness of the doctor during the study examinations.

The potential effects of the disease are not fully known, at this time, and may include long-term serious health consequences. In severe cases, this may result in hospitalization and/or death. Based on current knowledge from the Center for Disease Control (CDC), those at high-risk for severe illness from COVID-19 include older adults and people with underlying medical conditions.

During this study, all appropriate measures will be taken to minimize risks including the use of personal protective equipment such as masks and gloves, as well as proper sanitization. This is in conformance to guidance from the CDC, local health departments, and the state and county in which the study doctor's office is located. However, these measures may not completely eliminate the risks associated with contracting COVID-19.

If you are found to have contracted COVID-19 or feel ill with flu-like symptoms during participation in the study, you will not be permitted to continue in-office study follow-up visits but you will receive instructions and your condition will be monitored by the doctor and/or study staff.

#### 4.1.2 COVID-19 Risk Control Checklist:

Will include COVID-19 risk control methods that are required by a site to conduct JJVCI clinical studies. The risk controls are consistent with CDC, AOA, AAO Guidance. The Principle Investigator will review/sign the study specific checklist prior to the Site Initiation Meeting.

Study Number Site Number Principal Investigator (PI) Name

The following COVID-19 risk control methods are required to conduct Johnson & Johnson Vison Care clinical studies. Please review the following requirements and Initial each requirement.

| PI Initials | General Site Safety Planning Measures |
|---|---|
| ÷ | Signage within site describing Risk Control methods |
| 97 | Social Distancing practices throughout site (waiting rooms, lobby, exam rooms, etc.) |
| | Non-contact thermometer available to assess temperatures of staff and patients |
| Training on patient flow and physical distancing in waiting room Establish longer time frame between patient appointments to reduce persons in the site | |

| PI Initials | Site Staff Daily Safety Measures |
|---|---|
| As part of routine practice, site staff should regularly monitor themselves for fever and sympt of COVID-19, including temperature checks | |
| | Any staff member (including Investigators) showing signs of being sick or testing positive for COVID-19 should not be permitted to work and the Sponsor shall be informed NOTE: Inform JJVC in 24 hours of any significant impact to the study. |
| | Ensure that all staff wear a mask |


Title: Guidelines for COVID-19 Risk Mitigation

Document Type: Revision Number: 1

| Gloves should be required when working directly with patients and changed between each patient |
|---|
| Have staff thoroughly wash hands for at least 20 seconds or use an alcohol-based hand sanitizer when they arrive, before and after each patient, before eating and after using the bathroom. |
| Cleaning and disinfection procedures for exam rooms and instruments or equipment between patients with gloves. |
| Cleaning and disinfection procedures for commonly touched surfaces (doors, chairs, computers, phones, etc.) with gloves. |

| PI Initials | Before a Patient or Study Visit: |
|---|---|
| | Patients should be asked prior to entering the site about fever and respiratory illness and whether they or a family member have had contact with another person with confirmed COVID-19 in the past 2 to 14 days. Patients exhibiting signs of being sick should be rescheduled when their symptoms resolve. |
| | Instruct patients that companions should remain outside of the facility and not accompany the patient into the facility unless they are a parent/guardian of the patient or if they are a true caregiver and need to assist the patient |
| | Request the patient to call or text the office upon arrival so entrance to and movement through facility can be coordinated by site staff |

| PI Initials | Patients Entering the site: |
|---|---|
| the site All patients and companions must wear cloth or disposable mask Maintain social distancing. Waiting rooms or lobbies should be a | Temperature checks utilizing a non-contact thermometer for all patients and companions entering the site |
| | All patients and companions must wear cloth or disposable mask at all times in the site |
| | Maintain social distancing. Waiting rooms or lobbies should be as empty as possible. Advise seated patients to remain at least 6 feet from one another. |
| | Communal objects in (e.g. toys, reading materials, etc.) should be removed or cleaned regularly. |

I certify that I have read and agree to implement all the listed COVID-19 Risk Control Measures required for the conduct of Johnson & Johnson Vision Care studies.

Principal Investigator Signature and Date


Title: Guidelines for COVID-19 Risk Mitigation

Document Type: Revision Number: 1

#### RESOURCE LINKS

OSHA Training

https://www.osha.gov/SLTC/covid-19/controlprevention.html

Personal Protective Equipment (PPE) Training

CDC: https://www.cdc.gov/coronavirus/2019-ncov/hcp/using-ppe.html

I&R Training

ACUVUE® LensAssist: https://www.acuvue.com/lensassist

Clinic Preparedness Guides

CDC: https://www.cdc.gov/coronavirus/2019-ncov/hcp/clinic-preparedness html

AOA: https://aoa.uberflip.com/i/1240437-aoa-guidance-for-re-opening-practices-covid-19/1?m4=

American Optometric Association: <a href="https://www.aoa.org/optometry-practice-reactivation-preparedness-">https://www.aoa.org/optometry-practice-reactivation-preparedness-</a>

guide

In-Office Disinfection of Multi-Patient Use Diagnostic Contact Lenses
 https://www.gpli.info/wp-content/uploads/2020/03/2020-01-15-in-office-disinfecting-of-diagnostic-lenses.pdf

#### 4.1.3 Protocol Compliance Investigator(s) Signature Page:

Will include a statement indicating that the Principal Investigator (PI) agrees to conduct the study in compliance with all local, state, and governmental guidance's for COVID-19 risk mitigation.

I have read the suggested guidance provided by JJVCI pertaining to the COVID-19 risk mitigation, (COVID-19 Work Instruction in the Appendix of this protocol). I agree to conduct this study in compliance with local, state, governmental guidance for COVID-19 risks.

#### 4.1.4 Study Site Initiation Training Slides:

Will include suggestions to help mitigate potential transmission of COVID-19. Suggestions may include maintaining social distancing in the clinical site by staggered scheduling of study patients, wearing proper PPEs, frequent disinfection, and installing shields on the slit lamp and other applicable equipment.

#### 5.0 GUIDANCE FOR REMOTE SUBJECT VISITS

Potential disruptions to the study may be necessary due to current or future pandemic-related emergency restrictions. Possible disruption of the study as a result of COVID-19 control measures may lead to delays in scheduled follow-up visits.

Subjects may be delayed in being seen for study follow up visit(s), for example due to COVID-19 control measures or due to the subject's concerns or fears about COVID-19 risk. When appropriate, the remote assessment will be conducted to the extent possible. Discussions with the subject during remote assessments may include:


# Clinical Study Protocol Johnson & Johnson Vision Care, Inc. Guidelines for COVID-19 Risk Mitigation

| Title. | Guidennes for COVID-19 Risk Midgation | ducines for COVID-19 Risk Mitigation |
|---|---|---|
| Document Type: | | |
| Document Number | | Pavisian Number 1 |

| Procedure | Details |
|---|---|
| Subject Reported Ocular<br>Symptoms | Subjects will respond to a verbal open-ended symptoms questionnaire regarding the test article when applicable and feasible. |
| Change of Medical History<br>(Adverse Events) and<br>Concomitant Medications /<br>Therapies Review | Record any adverse events or medical history changes from the previous study visit with the subject/parents. Review the subject's concomitant medications/therapies and record any changes from the previous study visit. |
| Wearing Time and<br>Compliance | Record the average wearing time (including number of hours per day during weekdays and weekends, and number of days per week). Confirm compliance with the prescribed wear schedule. Record and discuss the lens wear compliance based on the subject's self-report. For example, the subjects will be asked the time of the day the subject typically puts on the study lenses in the morning and takes off in the evening, the number of days per week lenses were worn, and the number of consecutive days the subject didn't wear the study lenses, etc. |

The discussion with the subject will be documented in EDC under Tele-Visit and a minor protocol deviation will be noted. If during the telephone consultation, a subject states he/she wishes to discontinue participating in the study, instruct the subject to stop wearing the study lenses and schedule the subject to return to the clinic for a Final Evaluation at the at earliest possible time. Subjects should return all unused lenses to the clinic at the last visit.

Changes in study visit schedules, missed visits, or participant discontinuations may lead to missing data, including data related to protocol-specified procedures. Case report forms should capture specific information regarding the basis of missing data, including the relationship to the COVID-19 pandemic.

#### 6.0 STUDY CONDUCT DURING PANDEMIC

Title:

It is recognized that the Coronavirus Disease 2019 (COVID-19) pandemic may have an impact on the conduct of this clinical study due to, for example, self-isolation/quarantine by participants and study-site personnel; travel restrictions/limited access to public places, including Optometry Clinics; and changes in clinic procedures required to address the COVID-19 challenge.

Every effort should be made to adhere to protocol-specified assessments for study participants, including follow-up. However, if scheduled visits cannot be conducted in person at the study site it is suggested that assessments be performed to the extent possible remotely/virtually or delayed until such time that on-site visits can be resumed in order to continue participant monitoring in accordance with the protocol where possible. At each contact, participants will be interviewed to collect safety data. Key efficacy endpoint assessments should be performed if required and as feasible.

Modifications to protocol-required assessments may be permitted via COVID-19 Appendix after consultation with the participant, investigator, and the sponsor. Missed assessments/visits will be captured in the clinical trial management system for protocol deviations. Interruptions of test article wear or discontinuations of study interventions and withdrawal from the study should be documented with the prefix "COVID-19-related" in the case report form (CRF).


Title: Guidelines for COVID-19 Risk Mitigation

Document Type: Revision Number: 1

The sponsor will continue to monitor the conduct and progress of the clinical study, and any changes will be communicated to the sites and to the health authorities according to local guidance.

If a participant has tested positive for COVID-19, the investigator should contact the sponsor's responsible medical monitor to discuss initial plans for study intervention and follow-up. The medical monitor will notify the Safety Management Team of any subject(s) that have reported "COVID-19", "Asymptomatic COVID-19", or "Suspected COVID-19" adverse events within 24 hours of the notification.

Modifications made to the study conduct as a result of the COVID-19 pandemic will be summarized in the clinical study report.

COVID-19 screening procedures that may be mandated by local healthcare systems do not need to be reported as an amendment to the protocol even if done during clinical study visits.

#### 6.1 Monitoring Visits

When on-site monitoring by the sponsor is not feasible, the sponsor's site monitor will contact the study site to schedule remote visits. In such cases, on-site monitoring visits will resume when feasible, with increased frequency to address the source data verification backlog.

Even with staffing limitations during this COVID-19 pandemic, all routine operations related to clinical trials should be well-documented and archived as part of standard process. When conditions permit, all parties involved in this clinical trial should communicate relevant information in a timely manner so that all relevant parties remain sufficiently informed.

#### 6.1.1 Study Site Initiation:

During the period that this Work Instruction is in effect, Site Initiation Meetings and training of study site staff will be conducted remotely. The JJVCI study team will conduct training via Skype, Zoom, Microsoft Teams or similar software as well as utilize online training materials, as applicable. Study site training will be documented utilizing Site Initiation Report per Study Site Initiation

On-site visits may be considered when, for example, hands-on training or evaluation of site facilities is required. While on site, the Clinical Research Associate (CRA) will follow all local, state, and governmental policies for COVID-19 Risk Mitigation, including social distancing, wearing of PPE, etc. as applicable for the location of the study site.

#### 6.1.2 Interim Monitoring Visits (if applicable):

During the period that this Work Instruction is in effect, Interim Monitoring On-site visits will be kept to a minimum and include only those tasks that the CRA cannot perform remotely (e.g., source document verification, test article reconciliation, etc.).

To ensure data integrity during the conduct of all JJVC studies, clinical study teams will follow the study specific Clinical Monitoring Plan

While on site, the CRA will follow all local, state, and governmental policies for COVID-19 Risk Mitigation, including social distancing, wearing of PPE, etc. as applicable for the location of the study site.


Title: Guidelines for COVID-19 Risk Mitigation

Document Type: Revision Number: 1

#### 6.1.3 Study Site Closure:

During the period that this Work Instruction is in effect, the duration of the Study Site Closure Visit will be limited to tasks that the CRA cannot perform remotely (e.g., source document verification, test article final reconciliation and return, etc.).


Title: Guidelines for COVID-19 Risk Mitigation

Document Type: Revision Number: 1

Attachment A: Study Site Correspondence

XXXX XX, 2020

Re: COVID-19 Mitigation Plan, << CR-xxxx/protocol title>>

Dear << Principle Investigator>> and Study Team,

Coronavirus (COVID-19) has impacted several communities and business activities over the past several months. While we work toward the successful conduct of clinical studies, our commitment continues to be the safety of patients, healthcare professionals, and to our communities.

Therefore, we would like to share the following revisions/additions related to the above referenced Johnson & Johnson Vision Care company sponsored clinical trial(s) you are currently working on or considering participation within.

#### Protocol:

Guidelines for COVID-19 Risk Mitigation provided in the Appendix section.

#### **Protocol Signature Page:**

 Will include a statement indicating the Principle Investigator agrees to conduct the study in compliance with all local, state, and governmental guidelines for COVID-19 risk mitigation.

#### Informed Consent:

 Will include information concerning the study-associated risks related to the COVID-19 pandemic in bold font and/or boxed on the first page of the Informed consent document.

#### **COVID-19 Risk Control Checklist for Clinical Studies:**

 Will include COVID-19 risk control measures that are required to ensure the safety and health of subjects, site staff and monitors during the pandemic.

We want to encourage the need for open lines of communication about potential challenges you may foresee as the result of the current COVID-19 situation. Therefore, we encourage you to regularly connect with your respective Johnson & Johnson clinical study team (Clinical Research Associate (CRA), Lead CRA or Study Managers).

Thank you for your continued engagement, collaboration, and dedication to your study subjects during this challenging time.

Please file this letter in your site file study correspondence.


#### PROTOCOL COMPLIANCE INVESTIGATOR(S) SIGNATURE PAGE

Protocol Number and Title: CR-6371 Clinical Investigation of Visual Acuity in Contact Lens Wearers after Instillation of a Lipid-Based Eye Drop

Version and Date: 4.0 19 August 2020

I have read and understand the protocol specified above and agree on its content.

I agree to conduct this study according to ISO 14155,¹ GCP and ICH guidelines,² the Declaration of Helsinki,³ United States (US) Code of Federal Regulations (CFR),⁴ and the pertinent individual country laws/regulations and to comply with its obligations, subject to ethical and safety considerations. The Principal Investigator is responsible for ensuring that all clinical site personnel, including Sub-Investigators adhere to all ICH² regulations and GCP guidelines regarding clinical trials during and after study completion.

I will assure that no deviation from or changes to the protocol will take place without prior agreement from the Sponsor and documented approval from the Institutional Review Board (IRB), except where necessary to eliminate an immediate hazard(s) to the trial participants.

I am responsible for ensuring that all clinical site personnel including Sub-Investigators adhere to all ICH<sup>2</sup> regulations and GCP guidelines regarding clinical trials during and after study completion.

All clinical site personnel involved in the conduct of this study have completed Human Subjects Protection Training.

I agree to ensure that all clinical site personnel involved in the conduct of this study are informed about their obligations in meeting the above commitments.

I shall not disclose the information contained in this protocol or any results obtained from this study without written authorization.

I have read the suggested guidance provided by JJVCI pertaining to the COVID-19 risk mitigation, (COVID-19 Work Instruction in the Appendix of this protocol). I agree to conduct the study in compliance with all local, state, and governmental guidelines for COVID-19 risk mitigation.

| Principal Investigator: | | |
|-------------------------|------------------------------------------|------|
| | Signature | Date |
| | Name and Professional Position (Printed) | _ |
| Institution/Site: | | |
| | Institution/Site Name | |
| | Institution/Site Address | |
